CLINICAL TRIAL: NCT02299375
Title: A Study to Evaluate the Efficacy and Safety of 15mg BID Losmapimod (GW856553) Compared to Placebo in Frequently Exacerbating Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Safety and Efficacy Study of Losmapimod (GW856553) in Frequently Exacerbating Participants With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201496
Record Dates: First submitted 2014-11-03; First posted 2014-11-24 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Phase II clinical study; losmapimod; exacerbations; COPD; eosinophil sub-group
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losmapimod 15 mg (Experimental): Subjects with COPD will receive losmapimod 15 mg tablets orally, twice daily, approximately 12 hours apart and within 30 minutes after meals with a full glass of water for the duration of the treatment period in addition to standard of care, stratified according to whether a center collects sputum or not and current use of inhaled corticosteroid (ICS). Salbutamol metered dose inhaler (MDI) will be provided as a rescue medication.
  Interventions: Drug: Losmapimod tablets; Drug: Salbutamol MDI
- Placebo (Experimental): Subjects with COPD will receive placebo orally, twice daily, approximately 12 hours apart and within 30 minutes after meals with a full glass of water for the duration of the treatment period in addition to standard of care, stratified according to whether a center collects sputum or not and current use of ICS. Salbutamol MDI will be provided as a rescue medication.
  Interventions: Drug: Placebo tablets; Drug: Salbutamol MDI

INTERVENTIONS:
Drug: Losmapimod tablets — Losmapimod tablets will be provided as 15 mg strength in a formulation containing lactose. Administered orally, twice daily approximately 12 hours apart and with food and water for the duration of the treatment period. Participants will be instructed to take their medication with a full glass of water twice-daily within 30 minutes after meals for the duration of their treatment period.
  Arms: Losmapimod 15 mg
Drug: Placebo tablets — Placebo tablets will be provided in a formulation containing lactose and visually matching the losmapimod tablets. Administered orally, twice daily approximately 12 hours apart and with food and water for the duration of the treatment period. Participants will be instructed to take their medication with a full glass of water twice-daily within 30 minutes after meals for the duration of their treatment period
  Arms: Placebo
Drug: Salbutamol MDI — Salbutamol MDI will be provided as a rescue medication.

SUMMARY:
This is a randomised, double-blind, parallel-group, multi-centre study evaluating 15 milligram (mg) twice daily/ Bi-daily (BID) of losmapimod versus placebo, in addition to standard of care (SoC).

The primary objective of this study is to explore the therapeutic potential of losmapimod as a treatment to reduce the rate of exacerbations in the subset of participants with moderate-to-severe COPD who are at high risk of exacerbation, having experienced two or more moderate/severe exacerbations in the preceding 12 months, and who have <=2% of blood eosinophils at screening. As secondary objectives safety, effects on lung function, quality of life, pharmacokinetic (PK), biomarkers of both disease and inflammation shall be evaluated.

The duration of the treatment period is variable but will be at least 26 weeks and up to a maximum of 52 weeks, with the end of study date being established once the final participant has been randomized. The purpose of the variable dosing regimen is to enable participants to remain in the study for a longer duration, as it is anticipated that this will increase the likelihood of observing exacerbation events without increasing the overall study duration. It will also enable safety data on dosing periods beyond 6 months to be generated.

Approximately 200 participants in a 1:1 ratio between losmapimod and placebo will be randomized to the study. Sample size re-estimation will be performed during the course of the study to potentially increase the sample size up to a maximum of 600 participants.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis and severity: Participants with a clinical history of COPD (established by a physician) in accordance with the following definition by the American Thoracic Society/European Respiratory Society, for at least 6 months prior to enrolment. Participants must have evidence of airflow obstruction, defined as post-bronchodilator FEV1 equal to or less than 80% of predicted normal value calculated using "Third National Health and Nutrition Examination Survey" (NHANES III) reference equation at Visit 1 and a FEV1 / FVC ratio <=70% at Screening (Visit 1). Note: Post-bronchodilator spirometry will be performed approximately 10-15 minutes after the participants has self-administered 4 inhalations (i.e., total 400/360 [microgram] mcg) of salbutamol/albuterol via a Metered Dose Inhaler (MDI) (use of spacer will be optional). The study-provided central spirometry equipment will calculate the FEV1/FVC ratio and FEV1 percent predicted values.
* Exacerbation History: A documented history (e.g., medical record verification) in the 12 months prior to Visit 1 of >=2 COPD exacerbations resulting in prescription for antibiotics and/or oral corticosteroids or hospitalisation or extended observation in a hospital emergency room or outpatient centre. Note: Prior use of antibiotics alone does not qualify as a moderate exacerbation unless the use was specifically for the treatment of worsening symptoms of COPD.
* Existing COPD maintenance treatment: Participants must be receiving daily maintenance treatment for their COPD for at least 3 months prior to Screening. Notes: Participants receiving only "pro re nata" or as needed (PRN) COPD medications are not eligible for inclusion in the study. All participants will continue on their current Standard of Care (SoC) COPD medications throughout the entire duration of the study.
* Tobacco use: Participants with a current or prior history of >=10 pack-years of cigarette smoking at Screening (Visit 1). Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. One pack year =20 cigarettes smoked per day for 1 year or the equivalent. Number of pack years=(number of cigarettes per day/20) x number of years smoked.
* Sex: Male or female participants aged >=40 years at Screening (Visit 1). A female participant is eligible to participate if she is of non-child bearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli-international unit/milliliter (MIU/mL) and estradiol <40 picogram/milliliter (pg/mL) (<140 [Picomoles per liter] pmol/L) is confirmatory] or if of child-bearing potential is using a highly effective method for avoidance of pregnancy from 30 days before the first dose, for the duration of dosing and until 2 weeks post last-dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Corrected ECG QT interval (QTc)<450 milliseconds(msec) or QTc<480 msec for participants with bundle branch block. The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF), or another method, machine or manual over-read. For eligibility and withdrawal, ideally the same QT correction formula will be used for all participants. However, because this is not always possible, the same QT correction formula will be used for each individual participant to determine eligibility for and withdrawal from the study. The QTc will be based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period.

Exclusion Criteria:

* Eosinophils: >2.0% blood eosinophils at Screening (Visit 1)
* Concomitant medication: COPD Medication: Participants currently on chronic treatment with macrolides or Roflumilast; Long term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day. Oxygen PRN use (i.e. <=12 hours per day) is not exclusionary. Multidrug and toxin extrusion (MATE) transporter 1 (MATE1) inhibitors: cimetidine, pyrimethamine, trimethoprim (short course treatment with trimethoprim is allowed). Other medications: Chronic maintenance therapy with anti-Tumor Necrosis Factor (anti-TNF), anti-Interleukin-1 (anti-IL1), phosphodiesterase type 4 (PDE4) inhibitors, or any other immunosuppressive therapy (not including steroids) within 60 days prior to dosing. Any other investigational drug within 30 days or 5 half lives, whichever is longer prior to Screening Visit.
* Other respiratory disorders: Participants with asthma (as primary diagnosis) lung cancer, bronchiectasis, active sarcoidosis, active lung fibrosis, cystic fibrosis, idiopathic pulmonary hypertension, active interstitial lung diseases or other active pulmonary diseases. Participants with alpha-1-antitrypsin deficiency as the underlying cause of COPD.
* Participants with clinically significant sleep apnea who require use of continuous positive airway pressure (CPAP) device.
* Participants who require a non-invasive positive pressure ventilation (NIPPV) device (Note: Use of non invasive ventilation (NIV) in hospital as part of the medical management of an acute exacerbation is permitted.)
* Lung resection: Participants who have undergone previous lung reduction surgery (e.g. lobectomy, pneumonectomy, or lung volume reduction).
* COPD stability: Less than 30 days prior to Visit 1 have elapsed from completion of a course of antibiotics or oral corticosteroids for a recent COPD exacerbation.
* Evidence of pneumonia or a clinically significant abnormality not believed to be due to the presence of COPD on chest X-ray (posteroanterior with lateral) or computerised tomography (CT) scan (historic data up to 1 year may be used).
* Pulmonary rehabilitation program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Participants who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Alanine aminotransferase (ALT) >2x Upper limits of normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Malignancy: A current malignancy or previous history of cancer in remission for less than 12 months prior to Visit 1 (Participants that had localized carcinoma of the skin or cervix which was resected for cure will not be excluded).
* Other diseases/abnormalities: History or current evidence of clinically significant or uncontrolled cardiovascular, pulmonary, metabolic, neurological, endocrine (including uncontrolled diabetes or thyroid disease), renal, hepatic, haematological (including agranulocytosis) or gastrointestinal conditions that are uncontrolled on permitted therapy and in the opinion of the investigator and/or GSK Medical Monitor, places the participant at an unacceptable risk as participant in this trial or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study
* Viral infections: Presence of hepatitis B surface antigen (HBsAg), Hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. Note: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C Ribonucleic acid (RNA) polymerase chain reaction (PCR) test is obtained.
* A positive test for human immunodeficiency virus (HIV) antibody
* Tuberculosis (TB): Participant with active TB or who have previously tested positive for latent TB and not received treatment or prophylaxis following the positive test.
* Vaccination: Participants who have received live attenuated vaccines in the 6 weeks prior to randomization. The use of live attenuated vaccines during the treatment period and in the 4 weeks post-discontinuation of investigational product is prohibited.
* Drug/food allergy: Participants with a history of hypersensitivity to any of the study medications (e.g., lactose, magnesium stearate).
* Lactating females
* Pregnant females (as determined by positive urine human chorionic gonadotropin (hCG) test prior to dosing).
* Drug/alcohol abuse: Participants with a known or suspected history of alcohol or drug abuse within the last 2 years.
* Prior use of study medication/other investigational drugs: Participants who have received an investigational drug within 30 days of entry into this study or within 5 drug half-lives of the investigational drug, whichever is longer.
* Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participating in this study.
* Inability to read: In the opinion of the investigator, any participant who is unable to read and/or would not be able to complete study related materials.
* Non-compliance: Participants at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Questionable validity of consent: Participants with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- GSK Investigational Site, São Paulo, Brazil
- Bulgaria (3):
  - GSK Investigational Site, Dimitrovgrad
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Svoge
- Chile (3):
  - GSK Investigational Site, Talca, Maule Region
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Germany (8):
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Slovakia (5):
  - GSK Investigational Site, Humenné
  - GSK Investigational Site, Poprad
  - GSK Investigational Site, Spišská Nová Ves
  - GSK Investigational Site, Šaľa
  - GSK Investigational Site, Vráble
- South Korea (2):
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, (Barakaldo) Vizcaya
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobregat. Barcelona
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind (sponsor unblinded), parallel-group, multi-center study evaluating 15 milligrams (mg) twice daily (BID) of losmapimod versus placebo in addition to standard of care in male and female participants (par.) >=40 years of age having chronic obstructive pulmonary disease (COPD).
Pre-assignment Details: This study consisted of a 28 day screening period followed by treatment period (TP) of minimum 26 weeks. Total duration of TP was variable from 26 weeks to 52 weeks, and safety follow-up after 1 week. Total 365 par. were screened (175 par. failed), of which 190 par. passed screening and 184 par. were randomized in a TP.
Groups:
- Placebo: Participants with COPD received placebo orally, twice daily, approximately 12 hours apart and within 30 minutes after meals with a full glass of water for the duration of the treatment period in addition to standard of care, stratified according to whether a center collects sputum or not and current use of inhaled corticosteroid (ICS). Salbutamol metered dose inhaler (MDI) was provided as a rescue medication.
- Losmapimod 15 mg: Participants with COPD received losmapimod 15 mg tablets orally, twice daily, approximately 12 hours apart and within 30 minutes after meals with a full glass of water for the duration of the treatment period in addition to standard of care, stratified according to whether a center collects sputum or not and current use of ICS. Salbutamol MDI was provided as a rescue medication.
Period: Overall Study
Arm/Group | Placebo | Losmapimod 15 mg
Started | 94 | 90
Completed | 14 | 10
Not Completed | 80 | 80
Not completed — Adverse Event, serious fatal | 1 | 3
Not completed — Adverse Event, non-fatal | 8 | 9
Not completed — Lack of Efficacy | 1 | 3
Not completed — Protocol Violation | 1 | 3
Not completed — Other: Met stopping criteria | 1 | 0
Not completed — Other: Study closed/terminated | 66 | 55
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Losmapimod 15 mg | Total
Number analyzed (Participants) | 94 | 90 | 184
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (8.27) | 66.4 (6.66) | 65.5 (7.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 26 | 59
  Male | 61 | 64 | 125
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ Ethnicity: Japanese/East Asian /South East Asian Heritage | 10 | 9 | 19
  Race/ Ethnicity: White | 84 | 81 | 165

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Moderate and Severe Exacerbations of COPD
Description: An exacerbation of COPD, is defined as the worsening of 2 or more major symptoms (dyspnea, sputum volume, sputum purulence) or the worsening of any 1 major symptom together with any 1 of the minor symptoms (sore throat, cold, fever without other cause, increased cough and wheeze), for at least 2 consecutive days. Moderate-severe exacerbations were defined as use of antibiotics and/or oral steroids and/or hospitalization. Summary only included exacerbations for which a date of resolution or death was provided. Analysis was performed by using Bayesian inference assuming non-informative priors. The mean exacerbation rate was adjusted for treatment group, smoking status, ICS use and region. The adjusted posterior median was summarized per treatment group. The number of exacerbation events per participant was assumed to follow a negative binomial distribution. Modified Intent-to-Treat (mITT) Population comprised of all randomized par. who received at least one dose of study treatment.
Time Frame: From the start of the study treatment up to 53 Weeks
Population: mITT Population
Measure: Median (Standard Deviation); unit: Exacerbations per participant per year
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Exacerbations per participant per year | 0.84 (0.19) | 0.88 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; Adjusted median = 1.04, 95% CI 2-sided [0.63 to 1.73], Standard Deviation 0.28 — Data presented above are for 95% equal-tailed credible intervals. The estimated posterior probability that the true ratio losmapimod/placebo is <1 assuming noninformative priors is 0.44.The estimated posterior probability that the true ratio losmapi

2. Secondary Outcome: Time to First Occurrence of Moderate or Severe COPD Exacerbation
Description: The time to first moderate-severe COPD exacerbation in par. treated with losmapimod compared to placebo treated par. was evaluated. The time to the first on-treatment moderate-severe exacerbation was calculated as exacerbation onset date of first on-treatment exacerbation minus exposure start date plus 1. No statistical analysis was conducted. Data was summarized statistically only.
Time Frame: From the start of the study treatment up to 53 Weeks
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Days | 168.01 (106.222) | 160.18 (117.142)

3. Secondary Outcome: Number of Participants Having Any Adverse Events (AEs), Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinaemia were categorized as SAE. AEs were considered as on-treatment If AE onset date is on or after treatment start date & on or before treatment stop date. par. having any AE or SAE were included in analysis.
Time Frame: From the start of the study treatment up to 53 Weeks
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Participants
  Non-serious AEs | 34 | 38
  SAEs | 8 | 19

4. Secondary Outcome: Change From Baseline in Spirometry Parameters in Pre and Post Forced Expiratory Volume in 1 Second (FEV1); Pre and Post Forced Vital Capacity (FVC); Pre and Post Forced Expiratory Volume in 6 Seconds (FEV6).
Description: Pre and post FEV1, FVC and FEV6 were performed at Screening, Day 1 pre-dose and Weeks 2, 4, 8, 12, 18, 26, 39 and 52. Par. were asked to withheld all bronchodilator therapy included ipratropiumn bromide and salbutamol/albuterol for at least 4 hours prior to prebronchodilator spirometric test. Post-bronchodilator spirometric assessment was performed after inhalation of 400/360 micograms (µg) of salbutamol/albuterol in 10-15 minutes. Day 1 (pre-dose) values were considered as Baseline values. Change from Baseline was calculated as value at the indicated time point minus Baseline value. The maximum value of the 3 replicate assessments were used. Analysis performed using a mixed-effects repeated measures model. The adjusted mean values were summarized per treatment group. Par. were included in the analysis if they had at least one post-baseline measurement. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 52
Population: mITT Population
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Liters
  FEV1 pre-dose, Week 2, n = 90, 83: number analyzed (Participants) | 90 | 83
  FEV1 pre-dose, Week 2, n = 90, 83 | 0.002 (0.0241) | 0.028 (0.0258)
  FEV1 Pre-dose, Week 4, n=88, 82: number analyzed (Participants) | 88 | 82
  FEV1 Pre-dose, Week 4, n=88, 82 | -0.010 (0.0242) | 0.025 (0.0259)
  FEV1 Pre-dose, Week 8, n=81, 79: number analyzed (Participants) | 81 | 79
  FEV1 Pre-dose, Week 8, n=81, 79 | -0.031 (0.0247) | 0.028 (0.0261)
  FEV1 Pre-dose, Week 12, n=78, 71: number analyzed (Participants) | 78 | 71
  FEV1 Pre-dose, Week 12, n=78, 71 | -0.011 (0.0250) | -0.014 (0.0267)
  FEV1 Pre-dose, Week 18, n=67, 61: number analyzed (Participants) | 67 | 61
  FEV1 Pre-dose, Week 18, n=67, 61 | -0.037 (0.0260) | 0.013 (0.0277)
  FEV1 Pre-dose, Week 26, n=53, 52: number analyzed (Participants) | 53 | 52
  FEV1 Pre-dose, Week 26, n=53, 52 | -0.059 (0.0278) | 0.020 (0.0289)
  FEV1 Pre-dose, Week 39, n=28, 28: number analyzed (Participants) | 28 | 28
  FEV1 Pre-dose, Week 39, n=28, 28 | -0.085 (0.0342) | 0.001 (0.0353)
  FEV1 Pre-dose, Week 52, n=14, 11: number analyzed (Participants) | 14 | 11
  FEV1 Pre-dose, Week 52, n=14, 11 | -0.034 (0.0485) | 0.016 (0.0513)
  FEV1 post-dose, Week 2, n=89, 82: number analyzed (Participants) | 89 | 82
  FEV1 post-dose, Week 2, n=89, 82 | 0.012 (0.0188) | 0.026 (0.0203)
  FEV1 post-dose, Week 4, n=87, 81: number analyzed (Participants) | 87 | 81
  FEV1 post-dose, Week 4, n=87, 81 | -0.022 (0.0193) | 0.019 (0.0207)
  FEV1 post-dose, Week 8, n=80, 78: number analyzed (Participants) | 80 | 78
  FEV1 post-dose, Week 8, n=80, 78 | -0.010 (0.0232) | 0.023 (0.0242)
  FEV1 post-dose, Week 12, n=76, 69: number analyzed (Participants) | 76 | 69
  FEV1 post-dose, Week 12, n=76, 69 | -0.008 (0.0217) | -0.020 (0.0231)
  FEV1 post-dose, Week 18, n=66, 60: number analyzed (Participants) | 66 | 60
  FEV1 post-dose, Week 18, n=66, 60 | -0.035 (0.0256) | -0.012 (0.0271)
  FEV1 post-dose, Week 26, n=52, 51: number analyzed (Participants) | 52 | 51
  FEV1 post-dose, Week 26, n=52, 51 | -0.070 (0.0273) | 0.030 (0.0282)
  FEV1 post-dose, Week 39, n=27, 27: number analyzed (Participants) | 27 | 27
  FEV1 post-dose, Week 39, n=27, 27 | -0.086 (0.0346) | -0.031 (0.0356)
  FEV1 post-dose, Week 52, n=13, 10: number analyzed (Participants) | 13 | 10
  FEV1 post-dose, Week 52, n=13, 10 | -0.018 (0.0419) | 0.024 (0.0472)
  FEV6 pre-dose, Week 2, n = 90,82: number analyzed (Participants) | 90 | 82
  FEV6 pre-dose, Week 2, n = 90,82 | -0.007 (0.0353) | 0.045 (0.0381)
  FEV6 Pre-dose, Week 4, n=87, 81: number analyzed (Participants) | 87 | 81
  FEV6 Pre-dose, Week 4, n=87, 81 | -0.034 (0.0353) | 0.012 (0.0380)
  FEV6 Pre-dose, Week 8, n=81, 78: number analyzed (Participants) | 81 | 78
  FEV6 Pre-dose, Week 8, n=81, 78 | -0.043 (0.0400) | 0.032 (0.0424)
  FEV6 Pre-dose, Week 12, n=78, 71: number analyzed (Participants) | 78 | 71
  FEV6 Pre-dose, Week 12, n=78, 71 | -0.036 (0.0366) | -0.034 (0.0392)
  FEV6 Pre-dose, Week 18, n=67, 60: number analyzed (Participants) | 67 | 60
  FEV6 Pre-dose, Week 18, n=67, 60 | -0.073 (0.0413) | -0.014 (0.0441)
  FEV6 Pre-dose, Week 26, n=53, 52: number analyzed (Participants) | 53 | 52
  FEV6 Pre-dose, Week 26, n=53, 52 | -0.076 (0.0405) | -0.003 (0.0425)
  FEV6 Pre-dose, Week 39, n=28, 28: number analyzed (Participants) | 28 | 28
  FEV6 Pre-dose, Week 39, n=28, 28 | -0.102 (0.0486) | 0.013 (0.0507)
  FEV6 Pre-dose, Week 52, n=14, 11: number analyzed (Participants) | 14 | 11
  FEV6 Pre-dose, Week 52, n=14, 11 | -0.101 (0.0731) | 0.071 (0.0745)
  FEV6 post-dose, Week 2, n=89, 81: number analyzed (Participants) | 89 | 81
  FEV6 post-dose, Week 2, n=89, 81 | -0.003 (0.0296) | 0.023 (0.0319)
  FEV6 post-dose, Week 4, n=86, 80: number analyzed (Participants) | 86 | 80
  FEV6 post-dose, Week 4, n=86, 80 | -0.027 (0.0273) | 0.010 (0.0295)
  FEV6 post-dose, Week 8, n=80, 76: number analyzed (Participants) | 80 | 76
  FEV6 post-dose, Week 8, n=80, 76 | -0.039 (0.0313) | 0.012 (0.0331)
  FEV6 post-dose, Week 12, n=76, 69: number analyzed (Participants) | 76 | 69
  FEV6 post-dose, Week 12, n=76, 69 | -0.028 (0.0308) | -0.029 (0.0330)
  FEV6 post-dose, Week 18, n=66, 59: number analyzed (Participants) | 66 | 59
  FEV6 post-dose, Week 18, n=66, 59 | -0.060 (0.0367) | -0.035 (0.0392)
  FEV6 post-dose, Week 26, n=51, 51: number analyzed (Participants) | 51 | 51
  FEV6 post-dose, Week 26, n=51, 51 | -0.081 (0.0360) | 0.003 (0.0373)
  FEV6 post-dose, Week 39, n=27, 27: number analyzed (Participants) | 27 | 27
  FEV6 post-dose, Week 39, n=27, 27 | -0.095 (0.0428) | -0.067 (0.0443)
  FEV6 post-dose, Week 52, n=13, 10: number analyzed (Participants) | 13 | 10
  FEV6 post-dose, Week 52, n=13, 10 | -0.119 (0.0607) | -0.017 (0.0674)
  FVC, Pre-dose, Week 2, n =90, 83: number analyzed (Participants) | 90 | 83
  FVC, Pre-dose, Week 2, n =90, 83 | -0.018 (0.0389) | 0.038 (0.0417)
  FVC, Pre-dose, Week 4, n =88, 82: number analyzed (Participants) | 88 | 82
  FVC, Pre-dose, Week 4, n =88, 82 | -0.039 (0.0392) | 0.006 (0.0418)
  FVC, Pre-dose Week 8, n = 81, 79: number analyzed (Participants) | 81 | 79
  FVC, Pre-dose Week 8, n = 81, 79 | -0.061 (0.0401) | 0.011 (0.0422)
  FVC, Pre-dose, Week 12, n =78, 71: number analyzed (Participants) | 78 | 71
  FVC, Pre-dose, Week 12, n =78, 71 | -0.046 (0.0405) | -0.058 (0.0430)
  FVC, Pre-dose Week 18, n =67, 61: number analyzed (Participants) | 67 | 61
  FVC, Pre-dose Week 18, n =67, 61 | -0.093 (0.0422) | -0.021 (0.0447)
  FVC, Pre-dose Week 26, n=53, 52: number analyzed (Participants) | 53 | 52
  FVC, Pre-dose Week 26, n=53, 52 | -0.095 (0.0451) | -0.028 (0.0468)
  FVC, Pre-dose Week 39, n =28, 28: number analyzed (Participants) | 28 | 28
  FVC, Pre-dose Week 39, n =28, 28 | -0.115 (0.0558) | -0.033 (0.0574)
  FVC, Pre-dose Week 52, n =14, 11: number analyzed (Participants) | 14 | 11
  FVC, Pre-dose Week 52, n =14, 11 | -0.052 (0.0806) | 0.031 (0.0837)
  FVC, Post-dose Week 2, n =89, 82: number analyzed (Participants) | 89 | 82
  FVC, Post-dose Week 2, n =89, 82 | -0.007 (0.0359) | 0.037 (0.0385)
  FVC, Post-dose Week 4, n =87, 81: number analyzed (Participants) | 87 | 81
  FVC, Post-dose Week 4, n =87, 81 | -0.021 (0.0316) | 0.033 (0.0341)
  FVC, Post-dose Week 8, n =80, 78: number analyzed (Participants) | 80 | 78
  FVC, Post-dose Week 8, n =80, 78 | -0.052 (0.0366) | 0.019 (0.0385)
  FVC,Post-dose Week 12, n =76, 69: number analyzed (Participants) | 76 | 69
  FVC,Post-dose Week 12, n =76, 69 | -0.020 (0.0361) | -0.008 (0.0385)
  FVC, Post-dose Week 18, n =66, 60: number analyzed (Participants) | 66 | 60
  FVC, Post-dose Week 18, n =66, 60 | -0.075 (0.0422) | -0.016 (0.0449)
  FVC, Post-dose Week 26, n=52, 51: number analyzed (Participants) | 52 | 51
  FVC, Post-dose Week 26, n=52, 51 | -0.135 (0.0495) | 0.003 (0.0513)
  FVC, Post-dose Week 39, n =27, 27: number analyzed (Participants) | 27 | 27
  FVC, Post-dose Week 39, n =27, 27 | -0.092 (0.0499) | -0.043 (0.0518)
  FVC, Post-dose Week 52, n =13, 10: number analyzed (Participants) | 13 | 10
  FVC, Post-dose Week 52, n =13, 10 | -0.081 (0.0612) | -0.039 (0.0671)
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.371, MMRM — Analysis performed using a Mixed-effect Model Repeated Measures (MMRM) with covariates of treatment, smoking status at Screening, ICS use, region, Baseline, visit, treatment and Baseline by visit interactions. Toeplitz structure was used; Mean Difference (Net) = 0.026, 95% CI 2-sided [-0.031 to 0.084] — FEV1 pre-dose, Week 2
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.244, MMRM — Analysis performed using a Mixed-effect Repeated Measures model with covariates of treatment, smoking status at Screening, ICS use, region, Baseline, visit, treatment and Baseline by visit interactions. Toeplitz structure was used; Mean Difference (Net) = 0.035, 95% CI 2-sided [-0.024 to 0.093] — FEV1 pre-dose, Week 4
Statistical Analysis 3: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.050, MMRM — Analysis performed using a mixed-effects repeated measures model with covariates of treatment, smoking status at Screening, ICS use, region, Baseline, visit, treatment and Baseline by visit interactions. Toeplitz structure was used; Mean Difference (Net) = 0.059, 95% CI 2-sided [-0.000 to 0.119] — FEV1 pre-dose, Week 8
Statistical Analysis 4: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.942, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = -0.002, 95% CI 2-sided [-0.063 to 0.058] — FEV1 pre-dose, Week 12
Statistical Analysis 5: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.127, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.050, 95% CI 2-sided [-0.014 to 0.114] — FEV1 pre-dose, Week 18
Statistical Analysis 6: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.024, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.079, 95% CI 2-sided [0.011 to 0.148] — FEV1 pre-dose, Week 26
Statistical Analysis 7: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.057, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.086, 95% CI 2-sided [-0.003 to 0.174] — FEV1 pre-dose, Week 39
Statistical Analysis 8: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.481, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.050, 95% CI 2-sided [-0.090 to 0.191] — FEV1 pre-dose, Week 52
Statistical Analysis 9: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.521, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.014, 95% CI 2-sided [-0.030 to 0.059] — FEV1 post-dose, Week 2
Statistical Analysis 10: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.084, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.040, 95% CI 2-sided [-0.005 to 0.086] — FEV1 post-dose, Week 4
Statistical Analysis 11: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.266, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.033, 95% CI 2-sided [-0.025 to 0.090] — FEV1 post-dose, Week 8
Statistical Analysis 12: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.665, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = -0.012, 95% CI 2-sided [-0.066 to 0.042] — FEV1 post-dose, Week 12
Statistical Analysis 13: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.489, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.023, 95% CI 2-sided [-0.043 to 0.090] — FEV1 post-dose, Week 18
Statistical Analysis 14: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.007, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.099, 95% CI 2-sided [0.028 to 0.170] — FEV1 post-dose, Week 26
Statistical Analysis 15: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.248, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.055, 95% CI 2-sided [-0.039 to 0.148] — FEV1 post-dose, Week 39
Statistical Analysis 16: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.506, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.043, 95% CI 2-sided [-0.087 to 0.172] — FEV1 post-dose, Week 52
Statistical Analysis 17: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.223, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.051, 95% CI 2-sided [-0.032 to 0.134] — FEV6 pre-dose, Week 2
Statistical Analysis 18: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.276, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.046, 95% CI 2-sided [-0.037 to 0.129] — FEV6 pre-dose, Week 4
Statistical Analysis 19: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.131, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.075, 95% CI 2-sided [-0.023 to 0.173] — FEV6 pre-dose, Week 8
Statistical Analysis 20: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.949, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.003, 95% CI 2-sided [-0.084 to 0.090] — FEV6 pre-dose, Week 12
Statistical Analysis 21: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.259, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.059, 95% CI 2-sided [-0.044 to 0.163] — FEV6 pre-dose, Week 18
Statistical Analysis 22: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.152, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.073, 95% CI 2-sided [-0.027 to 0.172] — FEV6 pre-dose, Week 26
Statistical Analysis 23: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.076, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.114, 95% CI 2-sided [-0.012 to 0.241] — FEV6 pre-dose, Week 39
Statistical Analysis 24: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.107, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.171, 95% CI 2-sided [-0.038 to 0.381] — FEV6 pre-dose, Week 52
Statistical Analysis 25: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.484, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.025, 95% CI 2-sided [-0.046 to 0.097] — FEV6 post-dose, Week 2
Statistical Analysis 26: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.256, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.037, 95% CI 2-sided [-0.027 to 0.100] — FEV6 post-dose, Week 4
Statistical Analysis 27: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.184, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.052, 95% CI 2-sided [-0.025 to 0.128] — FEV6 post-dose, Week 8
Statistical Analysis 28: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.970, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = -0.001, 95% CI 2-sided [-0.077 to 0.074] — FEV6 post-dose, Week 12
Statistical Analysis 29: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.608, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.025, 95% CI 2-sided [-0.070 to 0.120] — FEV6 post-dose, Week 18
Statistical Analysis 30: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.071, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.084, 95% CI 2-sided [-0.007 to 0.175] — FEV6 post-dose, Week 26
Statistical Analysis 31: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.622, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.028, 95% CI 2-sided [-0.085 to 0.141] — FEV6 post-dose, Week 39
Statistical Analysis 32: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.277, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.102, 95% CI 2-sided [-0.086 to 0.291] — FEV6 post-dose, Week 52
Statistical Analysis 33: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.241, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.056, 95% CI 2-sided [-0.038 to 0.150] — FVC Pre-dose, Week 2
Statistical Analysis 34: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.348, MMRM; Mean Difference (Net) = 0.045, 95% CI 2-sided [-0.049 to 0.140] — FVC Pre-dose, Week 4
Statistical Analysis 35: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.138, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.073, 95% CI 2-sided [-0.024 to 0.169] — FVC Pre-dose, Week 8
Statistical Analysis 36: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.813, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = -0.012, 95% CI 2-sided [-0.111 to 0.087] — FVC Pre-dose, Week 12
Statistical Analysis 37: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.172, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.073, 95% CI 2-sided [-0.032 to 0.177] — FVC Pre-dose, Week 18
Statistical Analysis 38: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.242, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.067, 95% CI 2-sided [-0.045 to 0.180] — FVC Pre-dose, Week 26
Statistical Analysis 39: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.267, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.082, 95% CI 2-sided [-0.063 to 0.228] — FVC Pre-dose, Week 39
Statistical Analysis 40: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.471, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.083, 95% CI 2-sided [-0.143 to 0.309] — FVC Pre-dose, Week 52
Statistical Analysis 41: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.315, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.045, 95% CI 2-sided [-0.043 to 0.132] — FVC Post-dose, Week 2
Statistical Analysis 42: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.143, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.054, 95% CI 2-sided [-0.018 to 0.126] — FVC Post-dose, Week 4
Statistical Analysis 43: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.111, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.072, 95% CI 2-sided [-0.017 to 0.160] — FVC Post-dose, Week 8
Statistical Analysis 44: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.783, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.012, 95% CI 2-sided [-0.075 to 0.100] — FVC Post-dose, Week 12
Statistical Analysis 45: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.283, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.059, 95% CI 2-sided [-0.049 to 0.167] — FVC Post-dose, Week 18
Statistical Analysis 46: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.038, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.138, 95% CI 2-sided [0.008 to 0.267] — FVC Post-dose, Week 26
Statistical Analysis 47: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.467, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.048, 95% CI 2-sided [-0.083 to 0.180] — FVC Post-dose, Week 39
Statistical Analysis 48: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.640, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.042, 95% CI 2-sided [-0.138 to 0.222] — FVC Post-dose, Week 52

5. Secondary Outcome: Change From Baseline in Spirometry Parameters in Pre and Post FEV1/FVC, Percent Predicted (PP) FEV1, PP FEV6 and PP FVC
Description: Pre and post FEV1/FVC, PP FEV1, PP FEV6 and PP FVC were assessed at Screening, Day 1 pre-dose and Weeks 2, 4, 8, 12, 18, 26, 39 and 52. Par. were asked to withheld all bronchodilator therapy included ipratropiumn bromide and salbutamol/albuterol for at least 4 hours prior to the prebronchodilator spirometric test. Post-bronchodilator spirometric assessment was performed after inhalation of 400/360 µg of salbutamol/albuterol in 10-15 minutes. Day 1 (pre-dose) values were considered as Baseline values. Change from Baseline was calculated as value at indicated time point minus Baseline value. The maximum value of the 3 replicate assessments were used. Analysis performed using a mixed-effects repeated measures model. The adjusted mean values were summarized per treatment group. Par. were included in the analysis if they had at least one post-baseline measurement. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 52
Population: mITT Population.
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Percentage
  PP FVC, Week 2, n =90, 82: number analyzed (Participants) | 90 | 82
  PP FVC, Week 2, n =90, 82 | 0.72 (1.156) | 1.31 (1.228)
  PP FVC, Week 4, n =88, 81: number analyzed (Participants) | 88 | 81
  PP FVC, Week 4, n =88, 81 | -0.73 (1.160) | 1.72 (1.228)
  PP FVC, Week 8, n =81, 78: number analyzed (Participants) | 81 | 78
  PP FVC, Week 8, n =81, 78 | -2.05 (1.556) | 0.47 (1.604)
  PP FVC, Week 12 , n =78, 70: number analyzed (Participants) | 78 | 70
  PP FVC, Week 12 , n =78, 70 | -0.64 (1.324) | -0.78 (1.399)
  PP FVC, Week 18, n =67, 60: number analyzed (Participants) | 67 | 60
  PP FVC, Week 18, n =67, 60 | -1.58 (1.286) | 1.12 (1.356)
  PP FVC, Week 26, n =53, 51: number analyzed (Participants) | 53 | 51
  PP FVC, Week 26, n =53, 51 | -2.81 (1.518) | 1.88 (1.575)
  PP FVC, Week 39, n =28, 27: number analyzed (Participants) | 28 | 27
  PP FVC, Week 39, n =28, 27 | -2.06 (1.548) | 1.24 (1.604)
  PP FVC, Week 52, n =14, 11: number analyzed (Participants) | 14 | 11
  PP FVC, Week 52, n =14, 11 | -1.24 (2.017) | 0.92 (2.137)
  PP FEV1, Week 2, n =90, 82: number analyzed (Participants) | 90 | 82
  PP FEV1, Week 2, n =90, 82 | 0.28 (0.858) | 2.03 (0.932)
  PP FEV1, Week 4, n =88, 81: number analyzed (Participants) | 88 | 81
  PP FEV1, Week 4, n =88, 81 | -0.24 (0.877) | 1.52 (0.950)
  PP FEV1, Week 8, n =81, 78: number analyzed (Participants) | 81 | 78
  PP FEV1, Week 8, n =81, 78 | -1.14 (0.979) | 1.04 (1.037)
  PP FEV1, Week 12 , n =78, 70: number analyzed (Participants) | 78 | 70
  PP FEV1, Week 12 , n =78, 70 | -0.10 (0.940) | 0.12 (1.013)
  PP FEV1, Week 18, n =67, 60: number analyzed (Participants) | 67 | 60
  PP FEV1, Week 18, n =67, 60 | -0.79 (1.094) | 0.58 (1.172)
  PP FEV1, Week 26, n =53, 51: number analyzed (Participants) | 53 | 51
  PP FEV1, Week 26, n =53, 51 | -2.07 (1.075) | 1.26 (1.134)
  PP FEV1, Week 39, n =28, 27: number analyzed (Participants) | 28 | 27
  PP FEV1, Week 39, n =28, 27 | -2.33 (1.307) | 0.79 (1.370)
  PP FEV1, Week 52, n =14, 11: number analyzed (Participants) | 14 | 11
  PP FEV1, Week 52, n =14, 11 | -0.32 (1.714) | 2.03 (1.901)
  PP FEV6, Week 2, n =87, 75: number analyzed (Participants) | 87 | 75
  PP FEV6, Week 2, n =87, 75 | 0.63 (1.163) | 3.45 (1.252)
  PP FEV6, Week 4, n =84, 75: number analyzed (Participants) | 84 | 75
  PP FEV6, Week 4, n =84, 75 | -0.72 (1.135) | 2.15 (1.212)
  PP FEV6, Week 8, n =79, 74: number analyzed (Participants) | 79 | 74
  PP FEV6, Week 8, n =79, 74 | -1.71 (1.332) | 2.04 (1.395)
  PP FEV6, Week 12 , n =76, 67: number analyzed (Participants) | 76 | 67
  PP FEV6, Week 12 , n =76, 67 | -0.42 (1.214) | -0.02 (1.284)
  PP FEV6, Week 18, n =65, 56: number analyzed (Participants) | 65 | 56
  PP FEV6, Week 18, n =65, 56 | -1.47 (1.347) | 1.87 (1.438)
  PP FEV6, Week 26, n =51, 48: number analyzed (Participants) | 51 | 48
  PP FEV6, Week 26, n =51, 48 | -1.69 (1.359) | 1.84 (1.436)
  PP FEV6, Week 39, n =26, 24: number analyzed (Participants) | 26 | 24
  PP FEV6, Week 39, n =26, 24 | -2.10 (1.543) | 2.09 (1.652)
  PP FEV6, Week 52, n =13, 11: number analyzed (Participants) | 13 | 11
  PP FEV6, Week 52, n =13, 11 | 0.99 (2.936) | 3.66 (3.209)
  FEV1/FVC, Pre-dose, Week 2, n =90, 83: number analyzed (Participants) | 90 | 83
  FEV1/FVC, Pre-dose, Week 2, n =90, 83 | 0.22 (0.571) | 0.43 (0.611)
  FEV1/FVC, Pre-dose, Week 4, n =88, 82: number analyzed (Participants) | 88 | 82
  FEV1/FVC, Pre-dose, Week 4, n =88, 82 | 0.30 (0.674) | 0.43 (0.716)
  FEV1/FVC, Pre-dose Week 8, n = 81, 79: number analyzed (Participants) | 81 | 79
  FEV1/FVC, Pre-dose Week 8, n = 81, 79 | 0.10 (0.632) | 0.46 (0.663)
  FEV1/FVC, Pre-dose, Week 12, n =78, 71: number analyzed (Participants) | 78 | 71
  FEV1/FVC, Pre-dose, Week 12, n =78, 71 | 0.31 (0.649) | 0.02 (0.688)
  FEV1/FVC, Pre-dose Week 18, n =67, 61: number analyzed (Participants) | 67 | 61
  FEV1/FVC, Pre-dose Week 18, n =67, 61 | 0.11 (0.735) | 0.34 (0.780)
  FEV1/FVC, Pre dose Week 26, n=53, 52: number analyzed (Participants) | 53 | 52
  FEV1/FVC, Pre dose Week 26, n=53, 52 | -0.48 (0.767) | 0.84 (0.803)
  FEV1/FVC, Pre-dose Week 39, n =28, 28: number analyzed (Participants) | 28 | 28
  FEV1/FVC, Pre-dose Week 39, n =28, 28 | -1.36 (0.932) | 0.70 (0.963)
  FEV1/FVC, Pre-dose Week 52, n =14, 11: number analyzed (Participants) | 14 | 11
  FEV1/FVC, Pre-dose Week 52, n =14, 11 | -0.18 (1.177) | 1.26 (1.270)
  FEV1/FVC, Post-dose Week 2, n =89, 82: number analyzed (Participants) | 89 | 82
  FEV1/FVC, Post-dose Week 2, n =89, 82 | 0.09 (0.682) | 0.51 (0.726)
  FEV1/FVC, Post-dose Week 4, n =87, 81: number analyzed (Participants) | 87 | 81
  FEV1/FVC, Post-dose Week 4, n =87, 81 | -0.90 (0.619) | -0.23 (0.662)
  FEV1/FVC, Post-dose Week 8, n =80, 78: number analyzed (Participants) | 80 | 78
  FEV1/FVC, Post-dose Week 8, n =80, 78 | 0.12 (0.646) | 0.28 (0.679)
  FEV1/FVC,Post-dose Week 12, n =76, 69: number analyzed (Participants) | 76 | 69
  FEV1/FVC,Post-dose Week 12, n =76, 69 | -0.51 (0.693) | -0.97 (0.736)
  FEV1/FVC, Post-dose Week 18, n =66, 60: number analyzed (Participants) | 66 | 60
  FEV1/FVC, Post-dose Week 18, n =66, 60 | -0.65 (0.643) | -0.23 (0.682)
  FEV1/FVC, Post-dose Week 26, n=52, 51: number analyzed (Participants) | 52 | 51
  FEV1/FVC, Post-dose Week 26, n=52, 51 | -0.60 (2.272) | 3.23 (2.292)
  FEV1/FVC, Post-dose Week 39, n =27, 27: number analyzed (Participants) | 27 | 27
  FEV1/FVC, Post-dose Week 39, n =27, 27 | -1.27 (0.939) | 0.18 (0.961)
  FEV1/FVC, Post-dose Week 52, n =13, 10: number analyzed (Participants) | 13 | 10
  FEV1/FVC, Post-dose Week 52, n =13, 10 | 0.34 (1.280) | 1.51 (1.397)
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.661, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.60, 95% CI 2-sided [-2.08 to 3.27] — PP FVC, Week 2
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.074, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 2.44, 95% CI 2-sided [-0.24 to 5.12] — PP FVC, Week 6
Statistical Analysis 3: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.210, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 2.52, 95% CI 2-sided [-1.43 to 6.46] — PP FVC, Week 8
Statistical Analysis 4: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.933, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = -0.14, 95% CI 2-sided [-3.40 to 3.12] — PP FVC, Week 12
Statistical Analysis 5: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.091, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 2.70, 95% CI 2-sided [-0.43 to 5.82] — PP FVC, Week 18
Statistical Analysis 6: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.018, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 4.69, 95% CI 2-sided [0.82 to 8.56] — PP FVC, Week 26
Statistical Analysis 7: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.103, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 3.30, 95% CI 2-sided [-0.69 to 7.29] — PP FVC, Week 39
Statistical Analysis 8: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.448, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 2.16, 95% CI 2-sided [-3.50 to 7.82] — PP FVC, Week 52
Statistical Analysis 9: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.089, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 1.75, 95% CI 2-sided [-0.27 to 3.77] — PP FEV1, Week 2
Statistical Analysis 10: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.095, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 1.76, 95% CI 2-sided [-0.31 to 3.84] — PP FEV1, Week 4
Statistical Analysis 11: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.073, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 2.19, 95% CI 2-sided [-0.20 to 4.58] — PP FEV1, Week 8
Statistical Analysis 12: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.853, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.22, 95% CI 2-sided [-2.08 to 2.51] — PP FEV1, Week 12
Statistical Analysis 13: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.334, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 1.37, 95% CI 2-sided [-1.43 to 4.17] — PP FEV1, Week 18
Statistical Analysis 14: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.017, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 3.33, 95% CI 2-sided [0.61 to 6.05] — PP FEV1, Week 26
Statistical Analysis 15: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.077, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 3.13, 95% CI 2-sided [-0.34 to 6.59] — PP FEV1, Week 39
Statistical Analysis 16: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.355, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 2.34, 95% CI 2-sided [-2.70 to 7.38] — PP FEV1, Week 52
Statistical Analysis 17: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.044, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 2.82, 95% CI 2-sided [0.08 to 5.55] — PP FEV6, Week 2
Statistical Analysis 18: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.032, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 2.87, 95% CI 2-sided [0.25 to 5.49] — PP FEV6, Week 4
Statistical Analysis 19: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.025, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 3.75, 95% CI 2-sided [0.49 to 7.01] — PP FEV6, Week 8
Statistical Analysis 20: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.785, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.40, 95% CI 2-sided [-2.50 to 3.29] — PP FEV6, Week 12
Statistical Analysis 21: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.052, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 3.34, 95% CI 2-sided [-0.03 to 6.70] — PP FEV6, Week 18
Statistical Analysis 22: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.041, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 3.53, 95% CI 2-sided [0.14 to 6.92] — PP FEV6, Week 26
Statistical Analysis 23: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.043, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 4.19, 95% CI 2-sided [0.13 to 8.25] — PP FEV6, Week 39
Statistical Analysis 24: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.562, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 2.67, 95% CI 2-sided [-6.58 to 11.92] — PP FEV6, Week 52
Statistical Analysis 25: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.746, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.21, 95% CI 2-sided [-1.09 to 1.52] — Pre-dose FEV1/FVC, Week 2
Statistical Analysis 26: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.878, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.13, 95% CI 2-sided [-1.53 to 1.79] — Pre-dose FEV1/FVC, Week 4
Statistical Analysis 27: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.644, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.35, 95% CI 2-sided [-1.15 to 1.85] — Pre-dose FEV1/FVC, Week 8
Statistical Analysis 28: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.715, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = -0.29, 95% CI 2-sided [-1.86 to 1.28] — Pre-dose FEV1/FVC, Week 12
Statistical Analysis 29: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.803, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.24, 95% CI 2-sided [-1.62 to 2.10] — Pre-dose FEV1/FVC, Week 18
Statistical Analysis 30: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.184, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 1.32, 95% CI 2-sided [-0.63 to 3.27] — Pre-dose FEV1/FVC, Week 26
Statistical Analysis 31: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.102, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 2.05, 95% CI 2-sided [-0.42 to 4.52] — Pre-dose FEV1/FVC, Week 39
Statistical Analysis 32: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.383, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 1.44, 95% CI 2-sided [-1.85 to 4.73] — Pre-dose FEV1/FVC, Week 52
Statistical Analysis 33: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.607, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.43, 95% CI 2-sided [-1.20 to 2.06] — Post-dose FEV1/FVC, Week 2
Statistical Analysis 34: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.348, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.67, 95% CI 2-sided [-0.74 to 2.08] — Post-dose FEV1/FVC, Week 4
Statistical Analysis 35: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.826, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.17, 95% CI 2-sided [-1.32 to 1.65] — Post-dose FEV1/FVC, Week 8
Statistical Analysis 36: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.588, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = -0.46, 95% CI 2-sided [-2.13 to 1.21] — Post-dose FEV1/FVC, Week 12
Statistical Analysis 37: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.585, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 0.41, 95% CI 2-sided [-1.08 to 1.91] — Post-dose FEV1/FVC, Week 18
Statistical Analysis 38: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.231, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 3.82, 95% CI 2-sided [-2.48 to 10.12] — Post-dose FEV1/FVC, Week 26
Statistical Analysis 39: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.240, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 1.45, 95% CI 2-sided [-0.99 to 3.89] — Post-dose FEV1/FVC, Week 39
Statistical Analysis 40: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.517, MMRM — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Net) = 1.17, 95% CI 2-sided [-2.49 to 4.84] — Post-dose FEV1/FVC, Week 52

6. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Findings
Description: 12-lead ECGs were obtained in triplicate at Screening then singly at Baseline (day 1, pre-dose) and post dose at Weeks 2, 4, 8, 12, 26, 39, 52 and at follow up (Week 53) using an ECG machine that automatically calculates the heart rate (HR) and measures PR, QRS, QT, and QT duration corrected for heart rate by Fridericia's formula (QTcF) or QT duration corrected for heart rate by Bazett's formula (QTcB) intervals. Change in ECG findings were categorized as normal and abnormal. Abnormal ECG values could be clinically significant (CS) or not clinically significant (NCS), as determined by the investigator. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to 53 Weeks
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Participants
  Normal-SCREENING, (n=94,90) | 49 | 51
  Abnormal-NCS-SCREENING, (n=94,90) | 39 | 36
  Abnormal-CS-SCREENING, (n=94,90) | 9 | 5
  Normal-Baseline, (n=94,90) | 44 | 54
  Abnormal-NCS-Baseline, (n=94,90) | 46 | 31
  Abnormal-CS-Baseline, (n=94,90) | 4 | 5
  Normal-Week 2, (n=90,84): number analyzed (Participants) | 90 | 84
  Normal-Week 2, (n=90,84) | 40 | 52
  Abnormal-NCS-Week 2, (n=90,84): number analyzed (Participants) | 90 | 84
  Abnormal-NCS-Week 2, (n=90,84) | 45 | 29
  Abnormal-CS-Week 2, (n=90,84): number analyzed (Participants) | 90 | 84
  Abnormal-CS-Week 2, (n=90,84) | 5 | 3
  Normal-Week 4, (n=89,82): number analyzed (Participants) | 89 | 82
  Normal-Week 4, (n=89,82) | 45 | 53
  Abnormal-NCS-Week 4, (n=89,82): number analyzed (Participants) | 89 | 82
  Abnormal-NCS-Week 4, (n=89,82) | 40 | 27
  Abnormal-CS-Week 4, (n=89,82): number analyzed (Participants) | 89 | 82
  Abnormal-CS-Week 4, (n=89,82) | 4 | 2
  Normal-Week 8, (n=80,80): number analyzed (Participants) | 80 | 80
  Normal-Week 8, (n=80,80) | 42 | 50
  Abnormal-NCS-Week 8, (n=80,80): number analyzed (Participants) | 80 | 80
  Abnormal-NCS-Week 8, (n=80,80) | 35 | 28
  Abnormal-CS-Week 8, (n=80,80): number analyzed (Participants) | 80 | 80
  Abnormal-CS-Week 8, (n=80,80) | 3 | 2
  Normal-Week 12, (n=78,72): number analyzed (Participants) | 78 | 72
  Normal-Week 12, (n=78,72) | 45 | 42
  Abnormal-NCS-Week 12, (n=78,72): number analyzed (Participants) | 78 | 72
  Abnormal-NCS-Week 12, (n=78,72) | 29 | 29
  Abnormal-CS-Week 12, (n=78,72): number analyzed (Participants) | 78 | 72
  Abnormal-CS-Week 12, (n=78,72) | 4 | 1
  Normal-Week 26, (n=53,52): number analyzed (Participants) | 53 | 52
  Normal-Week 26, (n=53,52) | 31 | 35
  Abnormal-NCS-Week 26, (n=53,52): number analyzed (Participants) | 53 | 52
  Abnormal-NCS-Week 26, (n=53,52) | 21 | 16
  Abnormal-CS-Week 26, (n=53,52): number analyzed (Participants) | 53 | 52
  Abnormal-CS-Week 26, (n=53,52) | 1 | 1
  Normal-Week 39, (n=28,29): number analyzed (Participants) | 28 | 29
  Normal-Week 39, (n=28,29) | 18 | 20
  Abnormal-NCS-Week 39, (n=28,29): number analyzed (Participants) | 28 | 29
  Abnormal-NCS-Week 39, (n=28,29) | 9 | 8
  Abnormal-CS-Week 39, (n=28,29): number analyzed (Participants) | 28 | 29
  Abnormal-CS-Week 39, (n=28,29) | 1 | 1
  Normal-Week 52, (n=14,11): number analyzed (Participants) | 14 | 11
  Normal-Week 52, (n=14,11) | 11 | 7
  Abnormal-NCS-Week 52, (n=14,11): number analyzed (Participants) | 14 | 11
  Abnormal-NCS-Week 52, (n=14,11) | 2 | 4
  Abnormal-CS-Week 52, (n=14,11): number analyzed (Participants) | 14 | 11
  Abnormal-CS-Week 52, (n=14,11) | 1 | 0
  Normal-Follow up, (n=83,68): number analyzed (Participants) | 83 | 68
  Normal-Follow up, (n=83,68) | 37 | 42
  Abnormal-NCS-Follow up, (n=83,68): number analyzed (Participants) | 83 | 68
  Abnormal-NCS-Follow up, (n=83,68) | 40 | 25
  Abnormal-CS-Follow up, (n=83,68): number analyzed (Participants) | 83 | 68
  Abnormal-CS-Follow up, (n=83,68) | 6 | 1

7. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points
Description: SBP and DBP were taken at Screening, Baseline (day 1, pre-dose) and post dose at Weeks 2, 4, 8, 12, 26, 39, 52 and at follow up (Week 53). Measurements were taken in a semi-recumbent position after 5 minutes rest. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the value at day 1, pre-dose. Par. were included in the analysis if they had at least one post-baseline measurement. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Millimeter of mercury (mmHg)
  SBP, Week 2, (n=90,84): number analyzed (Participants) | 90 | 84
  SBP, Week 2, (n=90,84) | 0.2 (12.00) | -2.9 (11.85)
  SBP, Week 4, (n=89,82): number analyzed (Participants) | 89 | 82
  SBP, Week 4, (n=89,82) | -0.8 (11.49) | -0.4 (12.49)
  SBP, Week 8, (n=81,80): number analyzed (Participants) | 81 | 80
  SBP, Week 8, (n=81,80) | -1.9 (14.53) | -0.3 (11.48)
  SBP, Week 12, (n=78,72): number analyzed (Participants) | 78 | 72
  SBP, Week 12, (n=78,72) | 0.5 (12.97) | -1.6 (13.84)
  SBP, Week 26, (n=53,53): number analyzed (Participants) | 53 | 53
  SBP, Week 26, (n=53,53) | -1.5 (15.39) | -1.3 (13.25)
  SBP, Week 39, (n=28,29): number analyzed (Participants) | 28 | 29
  SBP, Week 39, (n=28,29) | 0.3 (16.30) | -3.4 (10.99)
  SBP, Week 52, (n=14,11): number analyzed (Participants) | 14 | 11
  SBP, Week 52, (n=14,11) | 6.1 (17.81) | -7.6 (12.89)
  SBP, Follow up, (n=83,68): number analyzed (Participants) | 83 | 68
  SBP, Follow up, (n=83,68) | 1.8 (14.46) | 0.2 (13.41)
  DBP, Week 2, (n=90,84): number analyzed (Participants) | 90 | 84
  DBP, Week 2, (n=90,84) | -0.0 (7.18) | -3.8 (9.81)
  DBP, Week 4, (n=89,82): number analyzed (Participants) | 89 | 82
  DBP, Week 4, (n=89,82) | -0.3 (8.57) | -2.2 (9.32)
  DBP, Week 8, (n=81,80): number analyzed (Participants) | 81 | 80
  DBP, Week 8, (n=81,80) | -1.4 (8.75) | -1.5 (7.92)
  DBP, Week 12, (n=78,72): number analyzed (Participants) | 78 | 72
  DBP, Week 12, (n=78,72) | 1.5 (9.79) | -1.5 (9.59)
  DBP, Week 26, (n=53,53): number analyzed (Participants) | 53 | 53
  DBP, Week 26, (n=53,53) | 0.9 (8.33) | -1.2 (7.87)
  DBP, Week 39, (n=28,29): number analyzed (Participants) | 28 | 29
  DBP, Week 39, (n=28,29) | -0.5 (10.40) | -1.9 (9.58)
  DBP, Week 52, (n=14,11): number analyzed (Participants) | 14 | 11
  DBP, Week 52, (n=14,11) | 3.4 (8.08) | -0.2 (8.46)
  DBP, Follow up, (n=83,68): number analyzed (Participants) | 83 | 68
  DBP, Follow up, (n=83,68) | 1.5 (10.57) | -1.7 (9.94)

8. Secondary Outcome: Change From Baseline in Heart Rate (HR) Values at the Indicated Time Points
Description: HR was assessed at Screening, Baseline (day 1, pre-dose) and post dose at Weeks 2, 4, 8, 12, 26, 39, 52 and at follow up (Week 53). Measurements were taken in a semi-recumbent position after 5 minutes rest. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the value at day 1, pre-dose. Par. were included in the analysis if they had at least one post-baseline measurement. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Beats per minute (bpm)
  HR, Week 2, (n=90,84): number analyzed (Participants) | 90 | 84
  HR, Week 2, (n=90,84) | 1.2 (7.99) | 1.5 (9.92)
  HR, Week 4, (n=89,82): number analyzed (Participants) | 89 | 82
  HR, Week 4, (n=89,82) | 1.4 (7.18) | 0.6 (8.72)
  HR, Week 8, (n=81,80): number analyzed (Participants) | 81 | 80
  HR, Week 8, (n=81,80) | 1.0 (8.39) | 1.6 (9.50)
  HR, Week 12, (n=78,72): number analyzed (Participants) | 78 | 72
  HR, Week 12, (n=78,72) | 3.3 (8.80) | 2.2 (8.89)
  HR, Week 26, (n=53,53): number analyzed (Participants) | 53 | 53
  HR, Week 26, (n=53,53) | 4.1 (10.99) | 1.8 (8.32)
  HR, Week 39, (n=28,29): number analyzed (Participants) | 28 | 29
  HR, Week 39, (n=28,29) | 3.3 (9.48) | 4.4 (12.64)
  HR, Week 52, (n=14,11): number analyzed (Participants) | 14 | 11
  HR, Week 52, (n=14,11) | 4.3 (9.55) | 1.3 (8.72)
  HR, Follow up, (n=83,68): number analyzed (Participants) | 83 | 68
  HR, Follow up, (n=83,68) | 3.6 (6.72) | 4.2 (10.99)

9. Secondary Outcome: Plasma Losmapimod Area Under the Plasma Concentration Time Curve (AUC) From Time Zero to the End of Dosing Interval (AUC[0-tau])
Description: Pharmacokinetics (PK) of losmapimod was evaluated in participants with COPD using PK samples collected at pre-dose at Week 2 and Week 12. At Week 26, a sample was collected at pre-dose and a second sample was collected at 2 hours post-dose. Par. of mITT population that provided at least one observed concentration data in this study were considered for PK analysis. Drug plasma concentration-time data were modelled by nonlinear mixed effects modelling. AUC[0-tau] (tau=12 hours) was estimated from the model.
Time Frame: Pre-dose at Weeks 2 and 12; pre-dose and at 2 hours post-dose at Week 26
Population: PK Population.
Measure: Geometric Mean (95% Confidence Interval); unit: hour (h)*nanogram (ng)/milliliter (mL)
Arm/Group | Losmapimod 15 mg
Number analyzed (Participants) | 85
hour (h)*nanogram (ng)/milliliter (mL) | 668.5 [361.7 to 1235.6]

10. Secondary Outcome: Plasma Losmapimod Maximum Concentration (Cmax) and Lowest Concentration (Ctrough) at Steady State
Description: Pharmacokinetics of losmapimod was evaluated in participants with COPD using PK samples collected at pre-dose at Week 2 and Week 12. At Week 26, a sample was collected at pre-dose and a second sample was collected at 2 hours post-dose. Par. of mITT population that provided at least one observed concentration data in this study were considered for PK analysis (represented by n=X, X in the category titles). Drug plasma concentration-time data were modelled by nonlinear mixed effects modelling to develop a Population PK model. Cmax and Ctrough were estimated from the PK model.
Time Frame: Pre-dose at Weeks 2 and 12; pre-dose and at 2 hours post-dose at Week 26
Population: PK Population.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/ mL
Arm/Group | Losmapimod 15 mg
Number analyzed (Participants) | 85
ng/ mL
  Cmax | 49.7 [17.6 to 140.5]
  Ctrough | 23.7 [12.9 to 43.3]

11. Secondary Outcome: Change From Baseline in Frequency of Short Acting Beta-agonist or Anti-cholinergic Use
Description: Use of short acting bronchodilators (short-acting beta2-agonists or short-acting anti-cholinergic) was allowed and was recorded in daily patient diary. It included inhaled short-acting beta2-agonists (e.g. Ipratropium bromide, salbutamol, Ipratropium/salbutamol (albuterol) combination product) and short-acting anti-cholinergics (e.g., ipratropium bromide3). Use of these medications was allowed throughout the study except 4 hours prior to and during each clinic visit. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Average number of puffs per 24 hours
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Average number of puffs per 24 hours
  Week 4; n=85, 82: number analyzed (Participants) | 85 | 82
  Week 4; n=85, 82 | -0.0029 (0.73616) | -0.0400 (0.93329)
  Week 8; n=79, 79: number analyzed (Participants) | 79 | 79
  Week 8; n=79, 79 | 0.1143 (0.77946) | -0.1473 (1.26462)
  Week 12; n=76, 70: number analyzed (Participants) | 76 | 70
  Week 12; n=76, 70 | 0.0904 (1.06920) | 0.0022 (1.10426)
  Week 18; n=65, 61: number analyzed (Participants) | 65 | 61
  Week 18; n=65, 61 | 0.3163 (1.26883) | 0.1489 (0.97966)
  Week 26; n=51, 53: number analyzed (Participants) | 51 | 53
  Week 26; n=51, 53 | 0.2725 (1.43462) | 0.2098 (1.25768)
  Week 39; n=27, 27: number analyzed (Participants) | 27 | 27
  Week 39; n=27, 27 | 0.7109 (1.61447) | 0.3418 (1.39346)
  Week 52; n=14, 10: number analyzed (Participants) | 14 | 10
  Week 52; n=14, 10 | 0.4368 (1.22619) | -0.2881 (0.98057)

12. Secondary Outcome: Change From Baseline in St Georges Respiratory Questionnaire (SGRQ) Total, SGRQ Symptoms Score, SGRQ Activity Score and SGRQ Impact Score Over Time
Description: SGRQ-C is a health related quality of life questionnaire consisting of 14 questions. SGRQ-C total score was calculated as 100 multiplied by summed weights from all positive items divided by sum of weights for all items in questionnaire. Components (Activity, Symptoms, Impacts) were calculated as 100 multiplied by summed weights from all positive items in that component divided by sum of weights for all items in that component. Score range for SGRQ-C total is 0-100. Maximum weights for Activity, Symptoms and Impacts component is 982.9, 566.2 and 1652.8 respectively. SGRQ-C was transformed to SGRQ for reporting. Higher scores indicate greater disease impact. Score at Day 1, pre-dose (Week 0) was considered as Baseline. Change from Baseline was calculated as score at indicated time point minus Baseline value. Only those par. with analyzable data at the given time points (represented by n=X, X in category titles) were included in analysis.
Time Frame: Baseline and up to Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Scores on a scale
  SGRQ Total, Week 12, (n=74, 71): number analyzed (Participants) | 74 | 71
  SGRQ Total, Week 12, (n=74, 71) | -0.75 (1.541) | -1.42 (1.638)
  SGRQ Total, Week 26, (n=50, 49): number analyzed (Participants) | 50 | 49
  SGRQ Total, Week 26, (n=50, 49) | -2.20 (1.833) | -1.31 (1.904)
  SGRQ Total, Week 39, (n=28, 28): number analyzed (Participants) | 28 | 28
  SGRQ Total, Week 39, (n=28, 28) | -0.37 (2.451) | -3.19 (2.502)
  SGRQ Total, Week 52, (n=14, 11): number analyzed (Participants) | 14 | 11
  SGRQ Total, Week 52, (n=14, 11) | -2.95 (2.769) | -3.43 (3.098)
  SGRQ Symptoms, Week 12, (n=78, 72): number analyzed (Participants) | 78 | 72
  SGRQ Symptoms, Week 12, (n=78, 72) | -2.41 (1.999) | -4.08 (2.115)
  SGRQ Symptoms, Week 26, (n=52, 52): number analyzed (Participants) | 52 | 52
  SGRQ Symptoms, Week 26, (n=52, 52) | -5.04 (2.264) | -4.30 (2.335)
  SGRQ Symptoms, Week 39, (n=28, 29): number analyzed (Participants) | 28 | 29
  SGRQ Symptoms, Week 39, (n=28, 29) | -4.61 (3.411) | -8.21 (3.370)
  SGRQ Symptoms, Week 52, (n=14, 11): number analyzed (Participants) | 14 | 11
  SGRQ Symptoms, Week 52, (n=14, 11) | -3.69 (3.990) | -11.67 (4.296)
  SGRQ Activity, Week 12, (n=77, 71): number analyzed (Participants) | 77 | 71
  SGRQ Activity, Week 12, (n=77, 71) | -0.08 (1.968) | 1.15 (2.097)
  SGRQ Activity, Week 26, (n=50, 49): number analyzed (Participants) | 50 | 49
  SGRQ Activity, Week 26, (n=50, 49) | -0.33 (2.217) | 0.70 (2.303)
  SGRQ Activity, Week 39, (n=28, 28): number analyzed (Participants) | 28 | 28
  SGRQ Activity, Week 39, (n=28, 28) | 1.41 (3.027) | -1.00 (3.095)
  SGRQ Activity, Week 52, (n=14, 11): number analyzed (Participants) | 14 | 11
  SGRQ Activity, Week 52, (n=14, 11) | -1.80 (3.308) | 2.59 (3.650)
  SGRQ Impact, Week 12, (n=75, 71): number analyzed (Participants) | 75 | 71
  SGRQ Impact, Week 12, (n=75, 71) | -0.53 (1.780) | -2.22 (1.893)
  SGRQ Impact, Week 26, (n=52, 50): number analyzed (Participants) | 52 | 50
  SGRQ Impact, Week 26, (n=52, 50) | -1.84 (2.169) | -2.19 (2.255)
  SGRQ Impact, Week 39, (n=28, 28): number analyzed (Participants) | 28 | 28
  SGRQ Impact, Week 39, (n=28, 28) | -0.59 (2.868) | -2.80 (2.931)
  SGRQ Impact, Week 52, (n=14, 11): number analyzed (Participants) | 14 | 11
  SGRQ Impact, Week 52, (n=14, 11) | -2.01 (3.693) | -3.31 (4.099)
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.706, Mixed Models Analysis — Analysis was performed using a mixed-effects repeated measures model with covariates of treatment, smoking status at Screening, ICS use, region, Baseline, visit, treatment by visit and Baseline by visit interactions; Mean Difference (Net) = -0.67, 95% CI 2-sided [-4.20 to 2.85] — SGRQ Total, Week 12
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.694, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = 0.89, 95% CI 2-sided [-3.58 to 5.36] — SGRQ Total, Week 26
Statistical Analysis 3: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.382, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -2.83, 95% CI 2-sided [-9.23 to 3.58] — SGRQ Total, Week 39
Statistical Analysis 4: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.903, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -0.49, 95% CI 2-sided [-8.54 to 7.57] — SGRQ Total, Week 52
Statistical Analysis 5: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.481, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -1.67, 95% CI 2-sided [-6.33 to 2.99] — SGRQ Symptoms, Week 12
Statistical Analysis 6: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.793, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = 0.73, 95% CI 2-sided [-4.79 to 6.25] — SGRQ Symptoms, Week 26
Statistical Analysis 7: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.421, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -3.60, 95% CI 2-sided [-12.45 to 5.26] — SGRQ Symptoms, Week 39
Statistical Analysis 8: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.162, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -7.98, 95% CI 2-sided [-19.35 to 3.40] — SGRQ Symptoms, Week 52
Statistical Analysis 9: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.592, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = 1.23, 95% CI 2-sided [-3.31 to 5.78] — SGRQ Activity, Week 12
Statistical Analysis 10: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.704, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = 1.03, 95% CI 2-sided [-4.31 to 6.36] — SGRQ Activity, Week 26
Statistical Analysis 11: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.546, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -2.41, 95% CI 2-sided [-10.32 to 5.50] — SGRQ Activity, Week 39
Statistical Analysis 12: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.350, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = 4.39, 95% CI 2-sided [-5.06 to 13.84] — SGRQ Activity, Week 52
Statistical Analysis 13: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.411, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -1.69, 95% CI 2-sided [-5.75 to 2.37] — SGRQ Impact, Week 12
Statistical Analysis 14: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.896, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -0.35, 95% CI 2-sided [-5.67 to 4.97] — SGRQ Impact, Week 26
Statistical Analysis 15: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.559, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -2.21, 95% CI 2-sided [-9.73 to 5.30] — SGRQ Impact, Week 39
Statistical Analysis 16: Comparison: Placebo vs Losmapimod 15 mg; Test type: Superiority or Other; p = 0.809, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -1.29, 95% CI 2-sided [-12.19 to 9.60] — SGRQ Impact, Week 52

13. Secondary Outcome: Number of Participants With Abnormal Liver Events During the Treatment Period
Description: Various liver chemistry parameters were monitored periodically to ensure the safety and tolerability of Losmapimod as compared to placebo. Study treatments were discontinued for par. if alanine aminotransferase (ALT) absolute >= 5xupper limit of normal (ULN) or; ALT >= 3xULN persists for >=4 Weeks or; ALT>=3x ULN and bilirubin >=2xULN or; ALT>=3x ULN and International normalized ratio (INR) >=1.5 or; ALT>=3x ULN and cannot be monitored weekly for 4 Weeks or; ALT>=3x ULN symptomatic.
Time Frame: Up to Week 53
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Participants | 0 | 0

14. Secondary Outcome: Change From Baseline in Hemoglobin, Total Protein, Albumin and Mean Corpuscle Hemoglobin Concentration (MCHC) at the Indicated Time Points
Description: Blood samples were collected at Baseline (Day 1, pre-dose) and at Weeks 2, 4, 8, 12, 18, 26, 39, 52 (or at early withdrawal) and follow up (Week 53) to evaluate hemoglobin, total protein, albumin and MCHC. Values obtained at Day 1, pre-dose (Week 0) were considered as Baseline values. Change from Baseline was calculated as laboratory test value obtained at indicated time point minus Baseline value. If post-dose value was missing for a particular assessment visit, then no derivation were performed and the change from Baseline were set to missing for that visit. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Gram (G)/Liter (L)
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Gram (G)/Liter (L)
  Hemoglobin, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Hemoglobin, Week 2 (n=85,82) | -0.3 (7.12) | 0.0 (4.86)
  Hemoglobin, Week 4 (n=87,80): number analyzed (Participants) | 87 | 80
  Hemoglobin, Week 4 (n=87,80) | -0.6 (7.01) | -1.0 (6.34)
  Hemoglobin, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Hemoglobin, Week 8 (n=80,77) | -0.9 (8.38) | -2.5 (6.93)
  Hemoglobin, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Hemoglobin, Week 12 (n=76,70) | -0.5 (7.61) | -1.4 (9.90)
  Hemoglobin, Week 18 (n=66,61): number analyzed (Participants) | 66 | 61
  Hemoglobin, Week 18 (n=66,61) | 0.1 (9.24) | -2.3 (9.66)
  Hemoglobin, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Hemoglobin, Week 26 (n=52,50) | -0.7 (9.27) | -2.9 (8.86)
  Hemoglobin, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Hemoglobin, Week 39 (n=28,29) | 0.0 (11.71) | -0.1 (10.09)
  Hemoglobin, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Hemoglobin, Week 52 (n=14,11) | 2.9 (8.43) | -1.8 (7.90)
  Hemoglobin, Follow up (n=80,67): number analyzed (Participants) | 80 | 67
  Hemoglobin, Follow up (n=80,67) | -0.2 (9.30) | -4.5 (9.42)
  Albumin, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Albumin, Week 2 (n=90,84) | -0.3 (2.23) | -0.6 (2.55)
  Albumin, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Albumin, Week 4 (n=88,81) | -0.5 (2.35) | -0.3 (2.28)
  Albumin, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Albumin, Week 8 (n=81,79) | -1.1 (2.43) | -1.2 (2.38)
  Albumin, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Albumin, Week 12 (n=78,72) | -0.4 (2.62) | -0.8 (2.64)
  Albumin, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Albumin, Week 18 (n=67,60) | -1.1 (2.53) | -1.1 (2.32)
  Albumin, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Albumin, Week 26 (n=53,50) | -0.9 (2.89) | -1.1 (2.25)
  Albumin, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Albumin, Week 39 (n=28,29) | -0.8 (2.76) | -1.2 (2.35)
  Albumin, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Albumin, Week 52 (n=14,11) | -0.4 (2.95) | -1.5 (2.07)
  Albumin, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Albumin, Follow up (n=80,68) | -0.8 (2.49) | -1.6 (2.71)
  Total protein, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Total protein, Week 2 (n=90,84) | -0.4 (3.68) | -1.6 (2.96)
  Total protein, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Total protein, Week 4 (n=88,81) | -0.8 (3.93) | -1.2 (3.18)
  Total protein, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Total protein, Week 8 (n=81,79) | -1.8 (3.67) | -2.0 (3.01)
  Total protein, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Total protein, Week 12 (n=78,72) | -0.6 (4.14) | -0.8 (3.45)
  Total protein, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Total protein, Week 18 (n=67,60) | -0.8 (4.00) | -1.5 (2.66)
  Total protein, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Total protein, Week 26 (n=53,50) | -0.5 (4.59) | -1.5 (3.70)
  Total protein, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Total protein, Week 39 (n=28,29) | -0.6 (4.50) | -2.2 (3.51)
  Total protein, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Total protein, Week 52 (n=14,11) | -0.8 (4.66) | -3.0 (3.66)
  Total protein, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Total protein, Follow up (n=80,68) | -1.6 (4.05) | -2.0 (3.87)
  MCHC, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  MCHC, Week 2 (n=85,82) | 0.1 (6.94) | 1.7 (6.40)
  MCHC, Week 4 (n=87,80): number analyzed (Participants) | 87 | 80
  MCHC, Week 4 (n=87,80) | 0.3 (6.31) | -0.6 (6.80)
  MCHC, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  MCHC, Week 8 (n=80,77) | -1.0 (7.63) | -0.9 (6.88)
  MCHC, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  MCHC, Week 12 (n=76,70) | -3.1 (8.45) | -3.3 (10.70)
  MCHC, Week 18 (n=66,61): number analyzed (Participants) | 66 | 61
  MCHC, Week 18 (n=66,61) | -5.0 (10.38) | -4.8 (8.75)
  MCHC, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  MCHC, Week 26 (n=52,50) | -4.4 (7.06) | -5.3 (8.48)
  MCHC, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  MCHC, Week 39 (n=28,29) | -2.8 (5.19) | -1.5 (5.35)
  MCHC, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  MCHC, Week 52 (n=14,11) | -3.9 (5.55) | -3.3 (6.15)
  MCHC, Follow up (n=80,67): number analyzed (Participants) | 80 | 67
  MCHC, Follow up (n=80,67) | 1.5 (9.77) | 0.6 (8.73)

15. Secondary Outcome: Change From Baseline in Hematocrit at the Indicated Time Points
Description: Blood samples were collected at Baseline (Day 1, pre-dose) and at Weeks 2, 4, 8, 12, 18, 26, 39, 52 (or at early withdrawal) and follow up (Week 53) to evaluate hematocrit. Values obtained at Day 1, pre-dose (Week 0) were considered as Baseline values. Change from Baseline was calculated as laboratory test value obtained at indicated time point minus Baseline value. If post-dose value was missing for a particular assessment visit, then no derivation were performed and the change from Baseline were set to missing for that visit. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
L
  Hematocrit, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Hematocrit, Week 2 (n=85,82) | -0.001 (0.0238) | -0.002 (0.0169)
  Hematocrit, Week 4 (n=87,80): number analyzed (Participants) | 87 | 80
  Hematocrit, Week 4 (n=87,80) | -0.002 (0.0236) | -0.002 (0.0218)
  Hematocrit, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Hematocrit, Week 8 (n=80,77) | -0.001 (0.0274) | -0.006 (0.0229)
  Hematocrit, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Hematocrit, Week 12 (n=76,70) | 0.002 (0.0251) | 0.000 (0.0361)
  Hematocrit, Week 18 (n=66,61): number analyzed (Participants) | 66 | 61
  Hematocrit, Week 18 (n=66,61) | 0.007 (0.0296) | -0.000 (0.0337)
  Hematocrit, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Hematocrit, Week 26 (n=52,50) | 0.003 (0.0302) | -0.000 (0.0318)
  Hematocrit, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Hematocrit, Week 39 (n=28,29) | 0.003 (0.0373) | 0.001 (0.0329)
  Hematocrit, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Hematocrit, Week 52 (n=14,11) | 0.014 (0.0231) | -0.001 (0.0255)
  Hematocrit, Follow up (n=80,67): number analyzed (Participants) | 80 | 67
  Hematocrit, Follow up (n=80,67) | -0.003 (0.0305) | -0.015 (0.0302)

16. Secondary Outcome: Change From Baseline in Absolute White Blood Cell (WBC) Count, Total Neutrophil, Total Lymphocyte, Basophil, Eosinophil, Monocyte and Platelet Count at the Indicated Time Point
Description: Blood samples were collected at Baseline (Day 1, pre-dose) and at Weeks 2, 4, 8, 12, 18, 26, 39, 52 (or at early withdrawal) and follow up (Week 53) to evaluate absolute WBC count, total neutrophil, total lymphocyte, basophil, absolute eosinophil, percentage eosinophil, monocyte and platelet count. Values obtained at Day 1, pre-dose (Week 0) were considered as Baseline values. Change from Baseline was calculated as laboratory test value obtained at the indicated time point minus Baseline value. If post-dose value was missing for a particular assessment visit, then no derivation were performed and the change from Baseline were set to missing for that visit. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Giga cells per liter (G/L)
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Giga cells per liter (G/L)
  Absolute WBC count, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Absolute WBC count, Week 2 (n=85,82) | -0.04 (1.586) | 0.21 (1.710)
  Absolute WBC count, Week 4 (n=86,80): number analyzed (Participants) | 86 | 80
  Absolute WBC count, Week 4 (n=86,80) | 0.03 (1.742) | 0.12 (2.116)
  Absolute WBC count, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Absolute WBC count, Week 8 (n=80,77) | 0.04 (1.474) | 0.32 (1.939)
  Absolute WBC count, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Absolute WBC count, Week 12 (n=76,70) | -0.07 (1.628) | 0.51 (1.905)
  Absolute WBC count, Week 18 (n=66,60): number analyzed (Participants) | 66 | 60
  Absolute WBC count, Week 18 (n=66,60) | 0.29 (1.921) | 0.17 (1.842)
  Absolute WBC count, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Absolute WBC count, Week 26 (n=52,50) | -0.07 (1.625) | 0.09 (1.876)
  Absolute WBC count, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Absolute WBC count, Week 39 (n=28,29) | 0.29 (1.777) | 1.08 (2.857)
  Absolute WBC count, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Absolute WBC count, Week 52 (n=14,11) | 0.86 (1.687) | 0.75 (1.637)
  Absolute WBC count, Follow up (n=79,67): number analyzed (Participants) | 79 | 67
  Absolute WBC count, Follow up (n=79,67) | 0.73 (1.691) | 0.50 (2.195)
  Total neutrophils, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Total neutrophils, Week 2 (n=85,82) | -0.038 (1.5980) | -0.080 (1.7982)
  Total neutrophils, Week 4 (n=86,80): number analyzed (Participants) | 86 | 80
  Total neutrophils, Week 4 (n=86,80) | -0.014 (1.7572) | -0.012 (2.0753)
  Total neutrophils, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Total neutrophils, Week 8 (n=80,77) | -0.052 (1.6060) | 0.060 (2.0525)
  Total neutrophils, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Total neutrophils, Week 12 (n=76,70) | 0.023 (1.7039) | 0.316 (2.0173)
  Total neutrophils, Week 18 (n=66,60): number analyzed (Participants) | 66 | 60
  Total neutrophils, Week 18 (n=66,60) | 0.189 (1.9556) | -0.161 (1.7378)
  Total neutrophils, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Total neutrophils, Week 26 (n=52,50) | -0.067 (1.4529) | -0.190 (1.8779)
  Total neutrophils, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Total neutrophils, Week 39 (n=28,29) | 0.240 (1.7846) | 0.689 (2.9389)
  Total neutrophils, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Total neutrophils, Week 52 (n=14,11) | 1.001 (1.8753) | 0.248 (1.4497)
  Total neutrophils, Follow up (n=79,67): number analyzed (Participants) | 79 | 67
  Total neutrophils, Follow up (n=79,67) | 0.555 (1.7317) | 0.309 (2.3168)
  Total lymphocyte, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Total lymphocyte, Week 2 (n=85,82) | 0.022 (0.4739) | 0.282 (0.7058)
  Total lymphocyte, Week 4 (n=86,80): number analyzed (Participants) | 86 | 80
  Total lymphocyte, Week 4 (n=86,80) | 0.043 (0.6599) | 0.161 (0.5497)
  Total lymphocyte, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Total lymphocyte, Week 8 (n=80,77) | 0.089 (0.5532) | 0.263 (0.7366)
  Total lymphocyte, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Total lymphocyte, Week 12 (n=76,70) | -0.083 (0.5983) | 0.210 (0.6986)
  Total lymphocyte, Week 18 (n=66,60): number analyzed (Participants) | 66 | 60
  Total lymphocyte, Week 18 (n=66,60) | 0.076 (0.4751) | 0.321 (0.6855)
  Total lymphocyte, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Total lymphocyte, Week 26 (n=52,50) | -0.042 (0.6673) | 0.296 (0.7236)
  Total lymphocyte, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Total lymphocyte, Week 39 (n=28,29) | 0.019 (0.4731) | 0.387 (0.6355)
  Total lymphocyte, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Total lymphocyte, Week 52 (n=14,11) | -0.107 (0.4707) | 0.449 (0.5762)
  Total lymphocyte, Follow up (n=79,67): number analyzed (Participants) | 79 | 67
  Total lymphocyte, Follow up (n=79,67) | 0.100 (0.5969) | 0.090 (0.6346)
  Basophils, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Basophils, Week 2 (n=85,82) | 0.000 (0.0194) | 0.002 (0.0290)
  Basophils, Week 4 (n=86,80): number analyzed (Participants) | 86 | 80
  Basophils, Week 4 (n=86,80) | -0.001 (0.0332) | -0.002 (0.0231)
  Basophils, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Basophils, Week 8 (n=80,77) | -0.003 (0.0288) | 0.003 (0.0254)
  Basophils, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Basophils, Week 12 (n=76,70) | 0.001 (0.0328) | 0.000 (0.0212)
  Basophils, Week 18 (n=66,60): number analyzed (Participants) | 66 | 60
  Basophils, Week 18 (n=66,60) | -0.002 (0.0249) | -0.002 (0.0191)
  Basophils, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Basophils, Week 26 (n=52,50) | 0.001 (0.0241) | -0.006 (0.0173)
  Basophils, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Basophils, Week 39 (n=28,29) | -0.001 (0.0180) | -0.005 (0.0190)
  Basophils, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Basophils, Week 52 (n=14,11) | -0.006 (0.0109) | -0.000 (0.0184)
  Basophils, Follow up (n=79,67): number analyzed (Participants) | 79 | 67
  Basophils, Follow up (n=79,67) | -0.004 (0.0305) | -0.000 (0.0234)
  Eosinophil, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Eosinophil, Week 2 (n=85,82) | 0.000 (0.0660) | 0.025 (0.0941)
  Eosinophil, Week 4 (n=86,80): number analyzed (Participants) | 86 | 80
  Eosinophil, Week 4 (n=86,80) | -0.002 (0.1092) | 0.013 (0.0713)
  Eosinophil, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Eosinophil, Week 8 (n=80,77) | 0.008 (0.0948) | 0.014 (0.0918)
  Eosinophil, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Eosinophil, Week 12 (n=76,70) | -0.001 (0.0817) | 0.013 (0.1173)
  Eosinophil, Week 18 (n=66,60): number analyzed (Participants) | 66 | 60
  Eosinophil, Week 18 (n=66,60) | 0.030 (0.1287) | 0.046 (0.1926)
  Eosinophil, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Eosinophil, Week 26 (n=52,50) | 0.037 (0.1554) | 0.051 (0.1646)
  Eosinophil, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Eosinophil, Week 39 (n=28,29) | 0.037 (0.0628) | 0.028 (0.1035)
  Eosinophil, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Eosinophil, Week 52 (n=14,11) | -0.001 (0.0539) | 0.006 (0.1688)
  Eosinophil, Follow up (n=79,67): number analyzed (Participants) | 79 | 67
  Eosinophil, Follow up (n=79,67) | 0.011 (0.0935) | 0.025 (0.0903)
  Monocytes, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Monocytes, Week 2 (n=85,82) | -0.029 (0.1598) | -0.024 (0.1898)
  Monocytes, Week 4 (n=86,80): number analyzed (Participants) | 86 | 80
  Monocytes, Week 4 (n=86,80) | 0.002 (0.1404) | -0.029 (0.1975)
  Monocytes, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Monocytes, Week 8 (n=80,77) | 0.001 (0.1785) | -0.014 (0.1653)
  Monocytes, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Monocytes, Week 12 (n=76,70) | -0.007 (0.1709) | -0.026 (0.2145)
  Monocytes, Week 18 (n=66,60): number analyzed (Participants) | 66 | 60
  Monocytes, Week 18 (n=66,60) | -0.010 (0.2023) | -0.025 (0.2235)
  Monocytes, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Monocytes, Week 26 (n=52,50) | 0.001 (0.2093) | -0.057 (0.1790)
  Monocytes, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Monocytes, Week 39 (n=28,29) | -0.005 (0.1210) | -0.020 (0.2376)
  Monocytes, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Monocytes, Week 52 (n=14,11) | -0.034 (0.1075) | 0.020 (0.1511)
  Monocytes, Follow up (n=79,67): number analyzed (Participants) | 79 | 67
  Monocytes, Follow up (n=79,67) | 0.071 (0.2319) | 0.083 (0.2190)
  Platelet count, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Platelet count, Week 2 (n=85,82) | -3.3 (45.84) | -2.3 (47.94)
  Platelet count, Week 4 (n=87,80): number analyzed (Participants) | 87 | 80
  Platelet count, Week 4 (n=87,80) | -6.4 (41.43) | -0.4 (35.50)
  Platelet count, Week 8 (n=79,77): number analyzed (Participants) | 79 | 77
  Platelet count, Week 8 (n=79,77) | -2.2 (40.51) | 6.3 (53.31)
  Platelet count, Week 12 (n=75,70): number analyzed (Participants) | 75 | 70
  Platelet count, Week 12 (n=75,70) | -10.0 (44.01) | 5.1 (55.82)
  Platelet count, Week 18 (n=66,59): number analyzed (Participants) | 66 | 59
  Platelet count, Week 18 (n=66,59) | 5.3 (53.14) | 3.2 (50.43)
  Platelet count, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Platelet count, Week 26 (n=52,50) | -2.7 (48.66) | -0.4 (42.21)
  Platelet count, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Platelet count, Week 39 (n=28,29) | -3.4 (35.47) | 0.0 (45.29)
  Platelet count, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Platelet count, Week 52 (n=14,11) | -13.6 (34.98) | -0.5 (30.06)
  Platelet count, Follow up (n=80,67): number analyzed (Participants) | 80 | 67
  Platelet count, Follow up (n=80,67) | 9.7 (58.86) | 10.5 (50.76)

17. Secondary Outcome: Change From Baseline in Eosinophil Percentage at the Indicated Time Points
Description: Blood samples were collected at Baseline (Day 1, pre-dose) and at Weeks 2, 4, 8, 12, 18, 26, 39, 52 (or at early withdrawal) and follow up (Week 53) to evaluate eosinophil percentage. Values obtained at Day 1, pre-dose (Week 0) were considered as Baseline values. Change from Baseline was calculated as laboratory test value obtained at the indicated time point minus Baseline value. If post-dose value was missing for a particular assessment visit, then no derivation were performed and the change from Baseline were set to missing for that visit. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Percent change
  Eosinophil percentage, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Eosinophil percentage, Week 2 (n=85,82) | 0.09 (0.969) | 0.30 (0.995)
  Eosinophil percentage, Week 4 (n=86,80): number analyzed (Participants) | 86 | 80
  Eosinophil percentage, Week 4 (n=86,80) | 0.03 (1.583) | 0.16 (0.930)
  Eosinophil percentage, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Eosinophil percentage, Week 8 (n=80,77) | 0.14 (1.419) | 0.11 (1.248)
  Eosinophil percentage, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Eosinophil percentage, Week 12 (n=76,70) | 0.08 (1.087) | 0.08 (1.517)
  Eosinophil percentage, Week 18 (n=66,60): number analyzed (Participants) | 66 | 60
  Eosinophil percentage, Week 18 (n=66,60) | 0.30 (1.513) | 0.60 (2.387)
  Eosinophil percentage, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Eosinophil percentage, Week 26 (n=52,50) | 0.58 (2.390) | 0.58 (2.082)
  Eosinophil percentage, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Eosinophil percentage, Week 39 (n=28,29) | 0.39 (0.865) | 0.21 (1.434)
  Eosinophil percentage, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Eosinophil percentage, Week 52 (n=14,11) | -0.11 (0.805) | 0.05 (2.819)
  Eosinophil percentage, Follow up (n=79,67): number analyzed (Participants) | 79 | 67
  Eosinophil percentage, Follow up (n=79,67) | -0.01 (1.245) | 0.29 (1.215)

18. Secondary Outcome: Change From Baseline in Total Bilirubin, Direct Bilirubin, Uric Acid and Creatinine at the Indicated Time Point
Description: Blood samples were collected at Baseline (Day 1, pre-dose) and at Weeks 2, 4, 8, 12, 18, 26, 39, 52 (or at early withdrawal) and follow up (Week 53) to evaluate total bilirubin, direct bilirubin, urice acid and creatinine. Values obtained at Day 1, pre-dose (Week 0) were considered as Baseline values. Change from Baseline was calculated as laboratory test value obtained at the indicated time point minus Baseline value. If post-dose value was missing for a particular assessment visit, then no derivation were performed and the change from Baseline were set to missing for that visit. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Micromole (UMOL)/ L
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Micromole (UMOL)/ L
  Total bilirubin, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Total bilirubin, Week 2 (n=90,84) | -0.5 (3.12) | 0.2 (3.62)
  Total bilirubin, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Total bilirubin, Week 4 (n=88,81) | 0.2 (3.07) | -0.1 (2.97)
  Total bilirubin, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Total bilirubin, Week 8 (n=81,79) | -0.4 (3.03) | -0.7 (3.28)
  Total bilirubin, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Total bilirubin, Week 12 (n=78,72) | -0.2 (3.33) | -0.1 (3.56)
  Total bilirubin, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Total bilirubin, Week 18 (n=67,60) | 0.0 (3.84) | 0.2 (2.66)
  Total bilirubin, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Total bilirubin, Week 26 (n=53,50) | 0.0 (3.03) | -0.5 (3.05)
  Total bilirubin, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Total bilirubin, Week 39 (n=28,29) | -0.0 (2.06) | 0.2 (3.55)
  Total bilirubin, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Total bilirubin, Week 52 (n=14,11) | 1.1 (3.38) | 0.9 (2.91)
  Total bilirubin, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Total bilirubin, Follow up (n=80,68) | 0.2 (3.62) | -0.4 (2.67)
  Direct bilirubin, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Direct bilirubin, Week 2 (n=90,84) | -0.1 (1.09) | 0.2 (1.04)
  Direct bilirubin, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Direct bilirubin, Week 4 (n=88,81) | 0.1 (0.89) | 0.0 (0.94)
  Direct bilirubin, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Direct bilirubin, Week 8 (n=81,79) | -0.0 (0.92) | -0.1 (0.98)
  Direct bilirubin, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Direct bilirubin, Week 12 (n=78,72) | 0.1 (0.92) | 0.3 (1.17)
  Direct bilirubin, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Direct bilirubin, Week 18 (n=67,60) | 0.1 (1.00) | 0.2 (0.98)
  Direct bilirubin, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Direct bilirubin, Week 26 (n=53,50) | -0.1 (0.79) | 0.0 (1.14)
  Direct bilirubin, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Direct bilirubin, Week 39 (n=28,29) | -0.1 (0.72) | 0.1 (0.88)
  Direct bilirubin, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Direct bilirubin, Week 52 (n=14,11) | -0.1 (1.14) | 0.1 (0.70)
  Direct bilirubin, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Direct bilirubin, Follow up (n=80,68) | 0.1 (1.09) | 0.0 (0.96)
  Uric acid, Week 2 (n=90,83): number analyzed (Participants) | 90 | 83
  Uric acid, Week 2 (n=90,83) | 1.7 (44.47) | -7.0 (45.87)
  Uric acid, Week 4 (n=88,80): number analyzed (Participants) | 88 | 80
  Uric acid, Week 4 (n=88,80) | -3.8 (53.43) | -14.0 (44.47)
  Uric acid, Week 8 (n=81,78): number analyzed (Participants) | 81 | 78
  Uric acid, Week 8 (n=81,78) | 2.1 (47.41) | -12.1 (52.91)
  Uric acid, Week 12 (n=78,71): number analyzed (Participants) | 78 | 71
  Uric acid, Week 12 (n=78,71) | 7.5 (54.68) | -10.2 (62.09)
  Uric acid, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Uric acid, Week 18 (n=67,60) | 6.7 (49.87) | -5.9 (54.33)
  Uric acid, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Uric acid, Week 26 (n=53,50) | 0.6 (54.09) | -3.7 (61.19)
  Uric acid, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Uric acid, Week 39 (n=28,29) | 13.7 (50.99) | 16.6 (87.59)
  Uric acid, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Uric acid, Week 52 (n=14,11) | 7.9 (48.23) | 8.3 (57.49)
  Uric acid, Follow up (n=80,67): number analyzed (Participants) | 80 | 67
  Uric acid, Follow up (n=80,67) | -2.6 (62.22) | 1.7 (63.56)
  Creatinine, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Creatinine, Week 2 (n=90,84) | 0.20 (7.974) | 3.22 (9.140)
  Creatinine, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Creatinine, Week 4 (n=88,81) | 0.04 (7.224) | 1.78 (9.899)
  Creatinine, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Creatinine, Week 8 (n=81,79) | 0.53 (11.111) | 2.23 (10.424)
  Creatinine, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Creatinine, Week 12 (n=78,72) | -0.11 (9.917) | 3.46 (17.547)
  Creatinine, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Creatinine, Week 18 (n=67,60) | 0.41 (11.973) | 5.32 (18.863)
  Creatinine, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Creatinine, Week 26 (n=53,50) | 1.61 (8.018) | 1.30 (8.927)
  Creatinine, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Creatinine, Week 39 (n=28,29) | 2.16 (6.164) | 5.64 (12.546)
  Creatinine, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Creatinine, Week 52 (n=14,11) | 2.94 (6.757) | 0.33 (5.150)
  Creatinine, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Creatinine, Follow up (n=80,68) | 0.62 (12.075) | 0.23 (9.463)

19. Secondary Outcome: Change From Baseline in Alanine Aminotransferase, Aspartate Aminotransferase, Alkaline Phosphatase and Gamma Glutamyl Transferase at the Indicated Time Points
Description: Blood samples were collected at Baseline (Day 1, pre-dose) and at Weeks 2, 4, 8, 12, 18, 26, 39, 52 (or at early withdrawal) and follow up (Week 53) to evaluate alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase and gamma glutamyl transferase at the indicated time point. Values obtained at Day 1, pre-dose (Week 0) were considered as Baseline values. Change from Baseline was calculated as laboratory test value obtained at the indicated time point minus Baseline value. If post-dose value was missing for a particular assessment visit, then no derivation were performed and the change from Baseline were set to missing for that visit. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: International units (IU)/ L
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
International units (IU)/ L
  Alanine aminotransferase, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Alanine aminotransferase, Week 2 (n=90,84) | -0.3 (3.78) | 1.2 (5.52)
  Alanine aminotransferase, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Alanine aminotransferase, Week 4 (n=88,81) | 1.8 (8.22) | 0.3 (6.56)
  Alanine aminotransferase, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Alanine aminotransferase, Week 8 (n=81,79) | -0.3 (6.00) | -0.1 (6.53)
  Alanine aminotransferase, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Alanine aminotransferase, Week 12 (n=78,72) | 1.3 (9.61) | 1.7 (7.48)
  Alanine aminotransferase, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Alanine aminotransferase, Week 18 (n=67,60) | 0.3 (8.03) | 2.4 (7.67)
  Alanine aminotransferase, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Alanine aminotransferase, Week 26 (n=53,50) | -0.2 (7.88) | 3.0 (10.79)
  Alanine aminotransferase, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Alanine aminotransferase, Week 39 (n=28,29) | 3.0 (14.98) | 1.9 (9.74)
  Alanine aminotransferase, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Alanine aminotransferase, Week 52 (n=14,11) | -1.1 (5.79) | 1.9 (3.24)
  Alanine aminotransferase, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Alanine aminotransferase, Follow up (n=80,68) | 0.7 (12.02) | 0.7 (6.86)
  Aspartate aminotransferase, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Aspartate aminotransferase, Week 2 (n=90,84) | -0.5 (3.68) | 1.4 (4.25)
  Aspartate aminotransferase, Week 4 (n=88,80): number analyzed (Participants) | 88 | 80
  Aspartate aminotransferase, Week 4 (n=88,80) | 2.0 (7.65) | 0.5 (5.16)
  Aspartate aminotransferase, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Aspartate aminotransferase, Week 8 (n=81,79) | -0.4 (6.54) | 0.5 (5.13)
  Aspartate aminotransferase, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Aspartate aminotransferase, Week 12 (n=78,72) | 2.2 (11.91) | 2.0 (7.73)
  Aspartate aminotransferase, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Aspartate aminotransferase, Week 18 (n=67,60) | 0.9 (5.72) | 2.9 (6.25)
  Aspartate aminotransferase, Week 26 (n=53,49): number analyzed (Participants) | 53 | 49
  Aspartate aminotransferase, Week 26 (n=53,49) | 0.3 (5.75) | 4.7 (9.94)
  Aspartate aminotransferase, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Aspartate aminotransferase, Week 39 (n=28,29) | 1.3 (6.50) | 2.4 (9.79)
  Aspartate aminotransferase, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Aspartate aminotransferase, Week 52 (n=14,11) | -1.1 (9.22) | 1.7 (3.23)
  Aspartate aminotransferase, Follow up (n=80,67): number analyzed (Participants) | 80 | 67
  Aspartate aminotransferase, Follow up (n=80,67) | 0.3 (6.55) | 0.1 (4.56)
  Alkaline phosphatase, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Alkaline phosphatase, Week 2 (n=90,84) | 0.3 (9.14) | -2.0 (11.62)
  Alkaline phosphatase, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Alkaline phosphatase, Week 4 (n=88,81) | 0.0 (10.43) | -2.8 (10.32)
  Alkaline phosphatase, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Alkaline phosphatase, Week 8 (n=81,79) | -2.5 (10.46) | -5.3 (12.71)
  Alkaline phosphatase, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Alkaline phosphatase, Week 12 (n=78,72) | -2.9 (12.67) | -4.7 (12.64)
  Alkaline phosphatase, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Alkaline phosphatase, Week 18 (n=67,60) | 1.0 (9.87) | -4.9 (13.57)
  Alkaline phosphatase, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Alkaline phosphatase, Week 26 (n=53,50) | 0.2 (13.06) | -4.4 (16.89)
  Alkaline phosphatase, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Alkaline phosphatase, Week 39 (n=28,29) | 0.9 (9.77) | -4.1 (22.29)
  Alkaline phosphatase, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Alkaline phosphatase, Week 52 (n=14,11) | 0.1 (6.39) | -9.5 (9.37)
  Alkaline phosphatase, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Alkaline phosphatase, Follow up (n=80,68) | -4.2 (15.26) | -4.4 (13.57)
  Gamma glutamyl transferase, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Gamma glutamyl transferase, Week 2 (n=90,84) | -0.3 (11.45) | -1.5 (16.55)
  Gamma glutamyl transferase, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Gamma glutamyl transferase, Week 4 (n=88,81) | 1.4 (19.82) | -3.7 (19.85)
  Gamma glutamyl transferase, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Gamma glutamyl transferase, Week 8 (n=81,79) | -1.8 (17.32) | -5.3 (20.20)
  Gamma glutamyl transferase, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Gamma glutamyl transferase, Week 12 (n=78,72) | -0.1 (17.11) | -1.1 (24.97)
  Gamma glutamyl transferase, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Gamma glutamyl transferase, Week 18 (n=67,60) | 0.6 (15.42) | -1.7 (21.15)
  Gamma glutamyl transferase, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Gamma glutamyl transferase, Week 26 (n=53,50) | -1.8 (13.53) | 2.5 (19.87)
  Gamma glutamyl transferase, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Gamma glutamyl transferase, Week 39 (n=28,29) | -1.7 (10.4) | 1.4 (25.46)
  Gamma glutamyl transferase, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Gamma glutamyl transferase, Week 52 (n=14,11) | -0.5 (13.39) | 0.1 (9.06)
  Gamma glutamyl transferase, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Gamma glutamyl transferase, Follow up (n=80,68) | -2.5 (17.16) | 0.1 (14.92)

20. Secondary Outcome: Change From Baseline in Chloride, Calcium, Glucose, Potassium, Sodium and Blood Urea Nitrogen at the Indicated Time Points
Description: Blood samples were collected at Baseline (Day 1, pre-dose) and at Weeks 2, 4, 8, 12, 18, 26, 39, 52 (or at early withdrawal) and follow up (Week 53) to evaluate calcium, chloride, glucose, potassium, sodium and blood urea nitrogenat the indicated time point. Values obtained at Day 1, pre-dose (Week 0) were considered as Baseline values. Change from Baseline was calculated as laboratory test value obtained at the indicated time point minus Baseline value. If post-dose value was missing for a particular assessment visit, then no derivation were performed and the change from Baseline were set to missing for that visit. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Millimole (MMOL)/L
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Millimole (MMOL)/L
  Chloride, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Chloride, Week 2 (n=90,84) | 0.3 (2.59) | 0.5 (2.40)
  Chloride, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Chloride, Week 4 (n=88,81) | -0.2 (2.42) | 1.1 (2.51)
  Chloride, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Chloride, Week 8 (n=81,79) | 0.3 (2.88) | 0.7 (2.85)
  Chloride, Week 12 (n=77,72): number analyzed (Participants) | 77 | 72
  Chloride, Week 12 (n=77,72) | 0.0 (2.48) | 0.2 (2.93)
  Chloride, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Chloride, Week 18 (n=67,60) | 0.2 (2.73) | 0.3 (2.66)
  Chloride, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Chloride, Week 26 (n=53,50) | -0.3 (3.35) | 0.5 (2.57)
  Chloride, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Chloride, Week 39 (n=28,29) | -0.8 (2.45) | 0.1 (2.15)
  Chloride, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Chloride, Week 52 (n=14,11) | -1.8 (2.12) | -1.4 (2.66)
  Chloride, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Chloride, Follow up (n=80,68) | -0.2 (2.87) | -0.5 (2.24)
  Calcium, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Calcium, Week 2 (n=90,84) | -0.002 (0.1031) | -0.042 (0.0774)
  Calcium, Week 4 (n=88,80): number analyzed (Participants) | 88 | 80
  Calcium, Week 4 (n=88,80) | -0.024 (0.1007) | -0.31 (0.0908)
  Calcium, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Calcium, Week 8 (n=81,79) | -0.017 (0.0934) | -0.039 (0.0843)
  Calcium, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Calcium, Week 12 (n=78,72) | -0.008 (0.1106) | -0.029 (0.0982)
  Calcium, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Calcium, Week 18 (n=67,60) | -0.017 (0.0891) | -0.033 (0.0928)
  Calcium, Week 26 (n=53,49): number analyzed (Participants) | 53 | 49
  Calcium, Week 26 (n=53,49) | -0.024 (0.0855) | -0.023 (0.1014)
  Calcium, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Calcium, Week 39 (n=28,29) | -0.017 (0.0922) | -0.032 (0.0927)
  Calcium, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Calcium, Week 52 (n=14,11) | 0.002 (0.1004) | -0.061 (0.0791)
  Calcium, Follow up (n=80,67): number analyzed (Participants) | 80 | 67
  Calcium, Follow up (n=80,67) | -0.018 (0.1042) | -0.010 (0.0959)
  Glucose, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Glucose, Week 2 (n=90,84) | -0.13 (1.456) | 0.22 (1.619)
  Glucose, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Glucose, Week 4 (n=88,81) | -0.01 (1.500) | 0.04 (1.204)
  Glucose, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Glucose, Week 8 (n=81,79) | 0.01 (1.330) | 0.28 (1.272)
  Glucose, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Glucose, Week 12 (n=78,72) | -0.08 (1.661) | 0.24 (1.439)
  Glucose, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Glucose, Week 18 (n=67,60) | 0.22 (1.607) | 0.50 (1.974)
  Glucose, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Glucose, Week 26 (n=53,50) | -0.08 (1.518) | 0.00 (1.117)
  Glucose, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Glucose, Week 39 (n=28,29) | -0.11 (1.553) | -0.16 (1.202)
  Glucose, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Glucose, Week 52 (n=14,11) | 0.31 (1.075) | -0.09 (0.896)
  Glucose, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Glucose, Follow up (n=80,68) | 0.20 (1.645) | 0.34 (2.104)
  Potassium, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Potassium, Week 2 (n=90,84) | 0.02 (0.349) | -0.01 (0.391)
  Potassium, Week 4 (n=88,80): number analyzed (Participants) | 88 | 80
  Potassium, Week 4 (n=88,80) | 0.01 (0.498) | 0.06 (0.393)
  Potassium, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Potassium, Week 8 (n=81,79) | 0.05 (0.406) | -0.03 (0.306)
  Potassium, Week 12 (n=77,72): number analyzed (Participants) | 77 | 72
  Potassium, Week 12 (n=77,72) | 0.02 (0.352) | -0.06 (0.354)
  Potassium, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Potassium, Week 18 (n=67,60) | 0.02 (0.390) | 0.14 (0.525)
  Potassium, Week 26 (n=53,49): number analyzed (Participants) | 53 | 49
  Potassium, Week 26 (n=53,49) | 0.02 (0.309) | -0.02 (0.381)
  Potassium, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Potassium, Week 39 (n=28,29) | 0.13 (0.395) | -0.03 (0.415)
  Potassium, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Potassium, Week 52 (n=14,11) | 0.10 (0.390) | -0.13 (0.422)
  Potassium, Follow up (n=80,67): number analyzed (Participants) | 80 | 67
  Potassium, Follow up (n=80,67) | 0.01 (0.385) | -0.02 (0.395)
  Sodium, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Sodium, Week 2 (n=90,84) | 0.1 (2.16) | -0.2 (2.06)
  Sodium, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Sodium, Week 4 (n=88,81) | -0.1 (2.18) | 0.3 (2.37)
  Sodium, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Sodium, Week 8 (n=81,79) | 0.0 (2.33) | -0.1 (2.50)
  Sodium, Week 12 (n=77,72): number analyzed (Participants) | 77 | 72
  Sodium, Week 12 (n=77,72) | -0.1 (1.96) | -0.4 (2.39)
  Sodium, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Sodium, Week 18 (n=67,60) | 0.1 (2.80) | -0.7 (2.49)
  Sodium, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Sodium, Week 26 (n=53,50) | 0.1 (2.92) | -0.2 (1.83)
  Sodium, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Sodium, Week 39 (n=28,29) | -0.4 (2.33) | -0.3 (2.18)
  Sodium, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Sodium, Week 52 (n=14,11) | -0.6 (1.28) | -0.9 (1.45)
  Sodium, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Sodium, Follow up (n=80,68) | -0.2 (2.40) | -0.1 (2.14)
  Blood urea nitrogen, Week 2 (n=90,84): number analyzed (Participants) | 90 | 84
  Blood urea nitrogen, Week 2 (n=90,84) | -0.04 (1.368) | 0.46 (1.474)
  Blood urea nitrogen, Week 4 (n=88,81): number analyzed (Participants) | 88 | 81
  Blood urea nitrogen, Week 4 (n=88,81) | -0.21 (1.399) | 0.14 (1.392)
  Blood urea nitrogen, Week 8 (n=81,79): number analyzed (Participants) | 81 | 79
  Blood urea nitrogen, Week 8 (n=81,79) | -0.11 (1.635) | 0.15 (1.464)
  Blood urea nitrogen, Week 12 (n=78,72): number analyzed (Participants) | 78 | 72
  Blood urea nitrogen, Week 12 (n=78,72) | -0.12 (1.511) | 0.62 (1.993)
  Blood urea nitrogen, Week 18 (n=67,60): number analyzed (Participants) | 67 | 60
  Blood urea nitrogen, Week 18 (n=67,60) | -0.41 (1.332) | 0.72 (2.310)
  Blood urea nitrogen, Week 26 (n=53,50): number analyzed (Participants) | 53 | 50
  Blood urea nitrogen, Week 26 (n=53,50) | -0.34 (1.267) | 0.24 (1.636)
  Blood urea nitrogen, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Blood urea nitrogen, Week 39 (n=28,29) | -0.26 (1.385) | 0.62 (1.680)
  Blood urea nitrogen, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Blood urea nitrogen, Week 52 (n=14,11) | 0.01 (0.975) | 1.07 (1.209)
  Blood urea nitrogen, Follow up (n=80,68): number analyzed (Participants) | 80 | 68
  Blood urea nitrogen, Follow up (n=80,68) | 0.07 (1.577) | 0.11 (1.545)

21. Secondary Outcome: Change From Baseline in Red Blood Cell Count at the Indicated Time Points
Description: Blood samples were collected at Baseline (Day 1, pre-dose) and at Weeks 2, 4, 8, 12, 18, 26, 39, 52 (or at early withdrawal) and follow up (Week 53) to evaluate Red blood cell count. Values obtained at Day 1, pre-dose (Week 0) were considered as Baseline values. Change from Baseline was calculated as laboratory test value obtained at the indicated time point minus Baseline value. If post-dose value was missing for a particular assessment visit, then no derivation were performed and the change from Baseline were set to missing for that visit. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Trillion cells per liter (TI/L)
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Trillion cells per liter (TI/L)
  Red blood cell count, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Red blood cell count, Week 2 (n=85,82) | -0.01 (0.248) | -0.00 (0.183)
  Red blood cell count, Week 4 (n=87,80): number analyzed (Participants) | 87 | 80
  Red blood cell count, Week 4 (n=87,80) | -0.03 (0.242) | -0.02 (0.219)
  Red blood cell count, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Red blood cell count, Week 8 (n=80,77) | -0.03 (0.281) | -0.05 (0.205)
  Red blood cell count, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Red blood cell count, Week 12 (n=76,70) | 0.02 (0.278) | 0.02 (0.328)
  Red blood cell count, Week 18 (n=66,61): number analyzed (Participants) | 66 | 61
  Red blood cell count, Week 18 (n=66,61) | 0.04 (0.341) | 0.00 (0.287)
  Red blood cell count, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Red blood cell count, Week 26 (n=52,50) | 0.01 (0.318) | -0.02 (0.268)
  Red blood cell count, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Red blood cell count, Week 39 (n=28,29) | 0.08 (0.352) | 0.09 (0.265)
  Red blood cell count, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Red blood cell count, Week 52 (n=14,11) | 0.23 (0.320) | 0.01 (0.230)
  Red blood cell count, Follow up (n=80,67): number analyzed (Participants) | 80 | 67
  Red blood cell count, Follow up (n=80,67) | 0.06 (0.354) | -0.04 (0.280)

22. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin at the Indicated Time Points
Description: Blood samples were collected at Baseline (Day 1, pre-dose) and at Weeks 2, 4, 8, 12, 18, 26, 39, 52 (or at early withdrawal) and follow up (Week 53) to evaluate mean corpuscle hemoglobin. Values obtained at Day 1, pre-dose (Week 0) were considered as Baseline values. Change from Baseline was calculated as laboratory test value obtained at the indicated time point minus Baseline value. If post-dose value was missing for a particular assessment visit, then no derivation were performed and the change from Baseline were set to missing for that visit. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Picograms
  Mean corpuscle hemoglobin, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Mean corpuscle hemoglobin, Week 2 (n=85,82) | 0.02 (0.551) | 0.03 (0.701)
  Mean corpuscle hemoglobin, Week 4 (n=87,80): number analyzed (Participants) | 87 | 80
  Mean corpuscle hemoglobin, Week 4 (n=87,80) | 0.09 (0.516) | -0.04 (0.480)
  Mean corpuscle hemoglobin, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Mean corpuscle hemoglobin, Week 8 (n=80,77) | 0.02 (0.801) | -0.20 (0.700)
  Mean corpuscle hemoglobin, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Mean corpuscle hemoglobin, Week 12 (n=76,70) | -0.22 (0.773) | -0.46 (0.964)
  Mean corpuscle hemoglobin, Week 18 (n=66,61): number analyzed (Participants) | 66 | 61
  Mean corpuscle hemoglobin, Week 18 (n=66,61) | -0.27 (1.167) | -0.52 (0.944)
  Mean corpuscle hemoglobin, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Mean corpuscle hemoglobin, Week 26 (n=52,50) | -0.25 (0.692) | -0.48 (0.983)
  Mean corpuscle hemoglobin, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Mean corpuscle hemoglobin, Week 39 (n=28,29) | -0.55 (1.121) | -0.60 (1.100)
  Mean corpuscle hemoglobin, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Mean corpuscle hemoglobin, Week 52 (n=14,11) | -0.72 (1.022) | -0.32 (0.676)
  Mean corpuscle hemoglobin, Follow up (n=80,67): number analyzed (Participants) | 80 | 67
  Mean corpuscle hemoglobin, Follow up (n=80,67) | -0.46 (1.130) | -0.73 (1.279)

23. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume at the Indicated Time Points
Description: Blood samples were collected at Baseline (Day 1, pre-dose) and at Weeks 2, 4, 8, 12, 18, 26, 39, 52 (or at early withdrawal) and follow up (Week 53) to evaluate mean corpuscle volume. Values obtained at Day 1, pre-dose (Week 0) were considered as Baseline values. Change from Baseline was calculated as laboratory test value obtained at the indicated time point minus Baseline value. If post-dose value was missing for a particular assessment visit, then no derivation were performed and the change from Baseline were set to missing for that visit. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 53
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | Losmapimod 15 mg
Number analyzed (Participants) | 94 | 90
Femtoliters
  Mean corpuscle volume, Week 2 (n=85,82): number analyzed (Participants) | 85 | 82
  Mean corpuscle volume, Week 2 (n=85,82) | 0.0 (1.72) | -0.4 (1.97)
  Mean corpuscle volume, Week 4 (n=87,80): number analyzed (Participants) | 87 | 80
  Mean corpuscle volume, Week 4 (n=87,80) | 0.1 (1.66) | 0.1 (1.88)
  Mean corpuscle volume, Week 8 (n=80,77): number analyzed (Participants) | 80 | 77
  Mean corpuscle volume, Week 8 (n=80,77) | 0.2 (2.49) | -0.4 (2.11)
  Mean corpuscle volume, Week 12 (n=76,70): number analyzed (Participants) | 76 | 70
  Mean corpuscle volume, Week 12 (n=76,70) | 0.3 (2.29) | -0.4 (2.45)
  Mean corpuscle volume, Week 18 (n=66,61): number analyzed (Participants) | 66 | 61
  Mean corpuscle volume, Week 18 (n=66,61) | 0.6 (2.85) | -0.1 (3.12)
  Mean corpuscle volume, Week 26 (n=52,50): number analyzed (Participants) | 52 | 50
  Mean corpuscle volume, Week 26 (n=52,50) | 0.5 (2.34) | 0.2 (3.07)
  Mean corpuscle volume, Week 39 (n=28,29): number analyzed (Participants) | 28 | 29
  Mean corpuscle volume, Week 39 (n=28,29) | -1.0 (3.50) | -1.4 (3.82)
  Mean corpuscle volume, Week 52 (n=14,11): number analyzed (Participants) | 14 | 11
  Mean corpuscle volume, Week 52 (n=14,11) | -1.4 (3.15) | 0.0 (2.05)
  Mean corpuscle volume, Follow up (n=80,67): number analyzed (Participants) | 80 | 67
  Mean corpuscle volume, Follow up (n=80,67) | -1.9 (2.73) | -2.4 (3.36)

ADVERSE EVENTS:
Time Frame: On-treatment SAEs and non-serious AEs were collected from start of Investigational Medicinal Product (Week 0) until Week 53 including 1 Week of follow up.
Description: On-treatment SAEs and non-serious AEs are reported for mITT Population, comprised of all par. who were randomized to treatment and who received at least one dose of study medication.
Groups:
- Losmapimod 15mg: Participants with COPD received losmapimod 15 mg tablets orally, twice daily, approximately 12 hours apart and within 30 minutes after meals with a full glass of water for the duration of the treatment period in addition to standard of care, stratified according to whether a center collects sputum or not and current use of ICS. Salbutamol MDI was provided as a rescue medication.
Arm/Group | Placebo | Losmapimod 15mg
All-Cause Mortality (participants affected / at risk) | 1/94 | 3/90
Serious Adverse Events (participants affected / at risk) | 8/94 | 19/90
Other Adverse Events (participants affected / at risk) | 9/94 | 13/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=94) | Losmapimod 15mg (N=90)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (9)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ileal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=94) | Losmapimod 15mg (N=90)
Nasopharyngitis (Infections and infestations) | 9 (13) | 13 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.